Sponsor: Insys Development Co, Inc.

Protocol Number: INS005-17-111

Statistical Analysis Plan

Date: 08Sep2017

# STATISTICAL ANALYSIS PLAN 08SEP2017 V1.0

A Phase 2, Randomized, Open Label, Multiple-Dose, Comparator, Parallel-Group, Safety and Tolerance Study of Buprenorphine Sublingual Spray (0.5 mg TID) versus Standard of Care Post-Operative Narcotic Therapy for the Treatment of Post-Operative Pain

#### Protocol Number: INS005-17-111 / NCT03254459

Protocol Version 1.0 (02AUG2017)

INS005-17-111 Admin Protocol Clarification Final 1.0 (10AUG2017)

INS005-17-111 Admin Protocol Clarification Final 2.0 (22AUG2017)

INS005-17-111 Admin Protocol Clarification Final 3.0 (30AUG2017)

INS005-17-111 Admin Protocol Clarification Final 4.0 (07SEP2017)

#### **SPONSORED BY**

Insys Development Company, Inc. 1333 South Spectrum Blvd, Suite 100 Chandler, AZ 85286

#### PREPARED BY



This document is confidential and proprietary to **Insys Development Company, Inc.**. Acceptance of this document constitutes agreement by the recipient that no unpublished information contained herein will be reproduced, published, or otherwise disclosed without the prior written approval of **Insys Development Company, Inc.**, except that this document may be disclosed to appropriate Institutional Review Boards under the condition that they keep the information confidential.

Sponsor: Insys Development Co, Inc. CONFIDENTIAL Statistical Analysis Plan

Protocol Number: INS005-17-111 Date: 08Sep2017

### DOCUMENT VERSION CONTROL

| Version Number | Date | Comments/Changes |
|---|---|---|
| V0.1 | 17AUG2017 | First Draft for Internal review |
| V0.2(S) | 22AUG2017 | First Draft for Sponsor review |
| V0.3(s) | 05SEP2017 | Incorporate sponsor comments, include Mock Shells for review |
| V1.0 | 08Sep2017 | Final v1.0 |

Sponsor: Insys Development Co, Inc.

Protocol Number: INS005-17-111

#### CONFIDENTIAL

Statistical Analysis Plan

Date: 08Sep2017

| | APPROVALS | |
|-----------|----------------------------------|----------------|
| Author: | | |
| | | Date: |
| Reviewed: | | 000 |
| | | SISEPSCU Date: |
| Approved | | |
| | Insys Development Company, Inc. | |
| Approved: | | |
| | In the David on mont Company Inc | Date: |
| | Insys Development Company, Inc. | |

Sponsor: Insys Development Co, Inc.

Protocol Number: INS005-17-111

CONFIDENTIAL

Statistical Analysis Plan

Date: 08Sep2017

### APPROVALS

| Author: | | |
|-----------|---------------------------------|-----------------------|
| | | 11 Sept 2017<br>Date: |
| Reviewed: | | |
| | | Date: |
| Approved | | 9/11/17 |
| | Insys Development Company, Inc. | |
| Approved: | Insys Development Company, Inc. | Date: |

| | APPROVALS | |
|-----------|---------------------------------|-------|
| Author: | | |
| | | Date: |
| Reviewed: | | |
| | | Date: |
| Approved | | |
| | Insys Development Company, Inc. | |
| Approved: | | |
| | Insys Development Company, Inc. | Date: |

Protocol Number: INS005-17-111

### TABLE OF CONTENTS

| LIS | T OF | IN-TEX | XT TABLES AND FIGURES | 7 |
|-----|------|--------|-------------------------------------------------|----|
| LIS | T OF | ABBR | EVIATIONS | 8 |
| 1. | PUR | POSE | OF THE ANALYSES | 10 |
| 2. | PRO | тосо | L SUMMARY | 11 |
| | 2.1 | Stud | dy Objectives | 11 |
| | 2 | 2.1.1 | Safety | 11 |
| | 2 | 2.1.2 | Efficacy | 11 |
| | 2.2 | Ove | rall Study Design and Plan | 11 |
| | 2.3 | Stud | dy Population | 13 |
| | 2.4 | Trea | atment Regimens | 14 |
| | 2 | 2.4.1 | Study Material | 14 |
| | 2 | 2.4.2 | Comparator Group | 14 |
| | 2.5 | Trea | atment Group Assignments or Randomization | 14 |
| | 2.6 | San | nple Size Determination | 15 |
| 3. | GEN | ERAL | ANALYSIS AND REPORTING CONVENTIONS | 16 |
| 4. | ANA | LYSIS | POPULATIONS | 18 |
| | 4.1 | Effic | cacy Population | 18 |
| | 4.2 | Safe | ety Population | 18 |
| | 4.3 | Disp | position of Subjects | 18 |
| | 4.4 | Maj | or Protocol Deviations | 18 |
| 5. | DEM | IOGRA | APHIC AND OTHER BASELINE CHARACTERISTICS | 19 |
| | 5.1 | Den | nographics and Baseline Characteristics | 19 |
| | 5.2 | Med | lical History | 19 |
| | 5.3 | Prio | r and Concomitant Medications/Surgeries Details | 19 |
| 6. | MEA | SURE | MENTS OF TREATMENT COMPLIANCE | 20 |
| | 6.1 | Stud | dy Medication Compliance | 20 |

Date: 08Sep2017

Protocol Number: INS005-17-111

| 7. | SAFE | ETY EVALUATION | 21 - |
|---|---|---|---|
| | 7.1 | Overview of Safety Analysis Methods | 21 - |
| | 7.2 | Adverse Events | 21 - |
| | 7.3 | Rescue Medication | 23 - |
| | 7.4 | Clinical Laboratory Evaluation | 24 - |
| | 7.5 | Vital Signs | 24 - |
| | 7.6 | Physical, Oral and ECG Exams | 25 - |
| | 7.7 | Serology Screens, Drug of Abuse and Alcohol Screens, Pregnancy T | est 25 |
| 8. | EFFIC | CACY EVALUATION | 26 - |
| 9. | OTHE | ER ANALYSES | 27 - |
| 10. | INTE | RIM ANALYSES AND DATA MONITORING | 28 - |
| 11. | CHAN | NGES TO THE ANALYSES PLANNED IN THE PROTOCOL | 29 - |
| 12. | REFE | ERENCES | 30 - |
| 13. | APPE | ENDICES | 31 - |
| | 13.1 | List of Tables for Final Study Report | 31 - |
| | 13.2 | List of Figures for Final Study Report | 33 - |
| | 13.3 | List of Listings for Final Study Report | 33 - |
| | 13.4 | TABLE, FIGURE AND LISTING SPECIFICATIONS | 36 |
| 14. | GENE | ERAL PROGRAMMING NOTES | 41 |
| | 14.1 | FIGURE SPECIFICATIONS | 69 |
| | 14.2 | LISTING SPECIFICATIONS | 70 |

| Sponsor: Insys | Development Co, Inc. | CONFIDENTIAL | Statistical Analysis Plan |
|---|---|---|---|
| Protocol Number: INS005-17-111 Date: 08Sep201 | | | |
| LIST OF IN | -TEXT TABLES AI | ND FIGURES | |
| Table 2-1 | Protocol-Specifie | d Visits and Visit Window | rs 13 - |
| Table 7-1 | Table of AE Start | Date Imputation Rules | 23 - |

Sponsor: Insys Development Co, Inc. CONFIDENTIAL Statistical Analysis Plan

Protocol Number: INS005-17-111 Date: 08Sep2017

#### LIST OF ABBREVIATIONS

ADaM Analysis Data Model

AE Adverse Event

ATC Anatomical Therapeutic Chemical

BMI Body Mass Index
BP Blood Pressure
CRF Case Report Form

CSR Clinical Study Report

ECG Electrocardiogram
ET Early Termination

HEENT Head, Ears, Eyes, Nose and Throat

HIV Human Immunovirus ICF Informed Consent Form

ICH International Conference on Harmonization

IP Investigational Product

IV Intra-Venous

IWRS Interactive Web Response System

MedDRA Medical Dictionary for Regulatory Activities

ODT Oral Dissolvable Tablet

PONV Post-Operative Nausea and Vomiting

PT Preferred Term
RTF Rich Text Format

SAE Serious Adverse Event/Experience

SAP Statistical Analysis Plan

SD Standard Deviation

SDTM Standard Data Table Model

SOC System Organ Class

TEAE Treatment Emergent Adverse Event

TID Three Times Per Day

Sponsor: Insys Development Co, Inc. CONFIDENTIAL Statistical Analysis Plan

Protocol Number: INS005-17-111 Date: 08Sep2017

WHO World Health Organization

Sponsor: Insys Development Co, Inc. Protocol Number: INS005-17-111 Date: 08Sep2017

#### 1. PURPOSE OF THE ANALYSES

This statistical analysis plan (SAP) is being developed after review of the Insys Development Company. Inc., protocol number INS005-17-111 Final Version 1.0, dated 02Aug2017 but before any analyses of the data. The SAP contains detailed information to aid in the performance of the statistical analysis and reporting of the study data for use in the final clinical study report (CSR). This SAP is being written with due consideration of the recommendations outlined in the most recent International Conference on Harmonization (ICH) E9 Guideline entitled Guidance for Industry: Statistical Principles for Clinical Trials and the most recent ICH E3 Guideline, entitled Guidance for Industry: Structure and Content of Clinical Study Reports and the most recent FDA draft Guidance for Industry - Analgesic Indications: Developing Drug and Biological Products, dated February 2014.

This SAP describes the data sets that will be analyzed and the subject characteristics, and safety assessments that will be evaluated. There will be no efficacy analysis in this study. This SAP provides details of the specific statistical methods that will be used. If additional analyses are required to supplement the planned analyses described in this SAP, they may be completed and will be identified in the CSR.

Sponsor: Insys Development Co, Inc.

Protocol Number: INS005-17-111 Date: 08Sep2017

#### 2. PROTOCOL SUMMARY

#### 2.1 Study Objectives

#### **2.1.1 Safety**

To evaluate the safety and tolerability based on the incidence of adverse experiences of Buprenorphine Sublingual Spray (0.5 mg three times daily [TID]) compared with standard post-operative narcotic therapy in subjects with postoperative pain. Standard post-operative narcotic therapy is defined as Morphine Intravenous Injection (IV) (4 mg TID) followed by Oxycodone Hydrochloride Tablet (10 mg TID).

#### 2.1.2 Efficacy

This is a safety and tolerability only study and so has no efficacy objectives.

#### 2.2 Overall Study Design and Plan

This is a Phase 2, randomized (stratified according to surgery and postoperative nausea and vomiting risk factors), open label, multiple-dose, comparator controlled, parallel-group, study to evaluate the safety and tolerability of Buprenorphine Sublingual Spray (0.5 mg TID) versus standard postoperative narcotic therapy in subjects with postoperative pain. Standard postoperative narcotic therapy is defined as Morphine IV (4 mg TID) for 24 hours followed by Oxycodone Hydrochloride Tablet (10 mg TID).

Subjects will be admitted to the study site on the morning of the scheduled surgery (Day 1), will remain at the study site until Postoperative Day 4 (a total of 3 nights at the study site) then be evaluated to participate in the outpatient setting and meet criteria in order to proceed to the outpatient treatment period Days 4 to 7. Subjects will subsequently return to the clinic for the Follow-up Visit on Day 8 (+2 day window). Subjects will be allowed rescue medication for pain and /or nausea at the investigator's discretion.

Screening Period: Subjects who meet all inclusion and no exclusion criteria will be eligible for enrollment. After providing written Informed Consent, subjects will undergo study specific screening procedures (please refer to the Protocol for complete list of procedures), including a review of inclusion and exclusion, demographics, medical history, concomitant medication use, assessment of postoperative nausea and vomiting (PONV) risk factors, physical and oral cavity examination, baseline laboratory testing, alcohol breath test, urine drug screening, HIV and hepatitis screening, 12-lead electrocardiogram (ECG), and pregnancy testing. Eligible subjects will complete all screening procedures within 28 days before the surgery (Days -28 to -1).

Statistical Analysis Plan

**Surgical Period:** On Day 1, anesthesia will be established using standardized techniques, as appropriate, for each surgical procedure. The surgical procedures will be either bunionectomy, breast augmentation, or abdominoplasty. For nausea prophylaxis, all subjects will receive a uniform standard of care regimen including 10 mg of dexamethasone at induction and 8 mg of ondansetron near the end of surgery. Vitals, pulse oximetry, and ECG measurements will be taken. Concomitant medications and Adverse Events will be recorded. Please refer to the Protocol for complete list of procedures.

Post-surgery and prior to randomization, subjects may be treated with intravenous morphine and or fentanyl for post-surgical analgesia (dose and frequency per the discretion of the investigator).

**Treatment Period - Inpatient**: After meeting post-surgical eligibility requirements and subsequently being randomized to treatment, subjects may receive their first dose of investigational drug any time between 0-4 hours after surgery. The first dose does not need to be immediately administered after meeting post-surgical eligibility requirements. Study medication administration after the first dose are to be administered every 8 hours (Treatment Period Days 1-7).

During the Treatment Period, approximately 100 subjects will be randomly assigned to 1 of 2 treatment groups: Buprenorphine Sublingual Spray 0.5 mg TID, or standard of care postoperative narcotic therapy. Randomization will be assigned by IWRS and stratified according to surgical procedure and baseline PONV risk factors. Vitals, pulse oximetry, and ECG measurements will be taken. Concomitant medications and Adverse Events will be recorded.

Pulse oximetry will be monitored continuously after surgery as a safety measure. An electrocardiogram (ECG) will be conducted after surgery but before the first dose of the study drug and serve as a baseline for comparison to subsequent tracings. The time of administration of the first dose of study drug will be defined as Time 0. The inpatient Treatment Period will continue through 72 hours after Time 0. Additional ECGs will be performed at 90 minutes, 12 hours, 24 hours, 48 hours and 72 hours after Time 0. Please refer to the Protocol for complete list of procedures.

**Treatment Period – Outpatient**: Investigators will determine if patients are able to proceed with the outpatient treatment period. After discharge to the outpatient portion of the trial, study drug will be administered by subjects at home according to the directions provided by study staff. Study personnel will dispense outpatient diary, study drug, and rescue medication for pain and nausea. Please refer to the Protocol for complete list of procedures.

Follow-up Visit on Day 8 (+2 day window): Subjects will be instructed to return any unused outpatient study drug to study personnel. Vitals, pulse oximetry, and ECG will be measured.

Sponsor: Insys Development Co, Inc. Protocol Number: INS005-17-111 Date: 08Sep2017

Concomitant medications and Adverse Events will be recorded. Subject outpatient diary will be collected and reviewed by study staff. Please refer to the Protocol for complete list of procedures.

Rescue medication: Rescue for inadequate analgesic response during confinement to the study center during the first 72 hours for pain will be acetaminophen 1000 mg every six hours and/or ketorolac 30 mg every six hours, as needed. On outpatient days 4-7 subjects will be provided with acetaminophen, and will be advised to take acetaminophen 1000 mg every six hours as needed for rescue analgesia.

Rescue for postoperative nausea during confinement to the study center during the first 72 hours will be Zofran 4 mg IV per the discretion of the clinician. On outpatient days 4-7, subjects will be provided with Zofran ODT (oral dissolvable tablet) to be taken as needed.

Subjects whose pain or nausea cannot be adequately managed (in the investigator's opinion) by a combination of study drug and rescue medication or who develop unacceptable side effects during the study will be discontinued from further study participation. Their pain or nausea will be managed according to usual standard of care at the investigator's discretion.

The protocol-defined visits are presented in the following table:

Table 2-1 **Protocol-Specified Visits and Visit Windows** 

| Study Phase | Visit Time |
|-------------------------------|---------------------|
| Screening | From days -28 to -1 |
| Surgical Period | Day 1 |
| Treatment Period - Inpatient | Days 1 to 4 |
| Treatment Period - Outpatient | Days 4 to 7 |
| Follow-up Visit | Day 8 (±2 days) |

#### Study Population

The study population will be males or females  $\ge 18$  and  $\le 65$  years of age, with body weight >45 kg and a body mass index (BMI) <40 kg/m2, and scheduled for elective bunionectomy, breast augmentation (in women only), or abdominoplasty.

Statistical Analysis Plan

Sponsor: Insys Development Co, Inc.

Protocol Number: INS005-17-111 Date: 08Sep2017

#### 2.4 Treatment Regimens

#### 2.4.1 Study Material

Buprenorphine Sublingual Spray, 0.5 mg TID manufactured for and supplied by Insys Development Company, Inc.

#### 2.4.2 Comparator Group

Morphine IV, 4 mg TID for 24 hrs, followed by Oxycodone Hydrochloride Tablet, 10 mg TID.

#### 2.5 Treatment Group Assignments or Randomization

Randomized treatment will be assigned utilizing a computer generated randomization scheme. Subjects who meet the inclusion criteria, do not fulfill any of the exclusion criteria and meet post-surgical eligibility requirements will be eligible for randomization into the study.

All study doses administered will be according to the IWRS specified treatment to ensure that study personnel will not be aware of the next subject's treatment assignment before the decision to randomize that subject has been made. The IWRS randomization algorithm will be such that the subjects will be stratified by surgical procedure and baseline PONV risk factors and randomly assigned to treatment administered in a 1:1 assignment ratio within the stratification categories. PONV risk will be assessed at screening to assess the likelihood of nausea and vomiting after surgery using the Apfel scale

| (PONV) Risk Factor | Points |
|----------------------------|--------|
| Assessment Risk Factors | |
| Post-operative Opioids (if | 1 |
| planned) | |
| Non Smoker | 1 |
| Female Gender | 1 |
| History of postoperative | 1 |
| nausea and vomiting / | |
| Motion Sickness | |
| Risk score = sum | 04 |

Patients with PONV risk factors of 0-2 will be stratified as low risk and 3-4 as high risk.

### 2.6 Sample Size Determination

No formal sample size estimate has been completed. A sample size of 50 subjects per treatment group is expected to be sufficient to achieve the study objectives.

Statistical Analysis Plan

Sponsor: Insys Development Co, Inc. CONFIDENTIAL

Protocol Number: INS005-17-111 Date: 08Sep2017

#### 3. GENERAL ANALYSIS AND REPORTING CONVENTIONS

This section discusses general policies to be employed in the analysis and reporting of the data from the study. Departures from these general policies are provided in the specific detailed sections of this SAP. When this situation occurs, the rules set forth in the specific section take precedence over the general policies.

All continuous study assessments will be summarized by treatment and time point (as applicable) using descriptive statistics (n, mean, SD, median, minimum, and maximum). All of the categorical study assessments will be summarized by treatment and time point (as applicable) using frequency counts and percentages. Changes from baseline for continuous outcomes will be presented as their corresponding continuous measures for post-baseline visits. All relevant study data will be listed by treatment group, subject, and time point (as applicable).

No preliminary rounding will be performed; rounding will only occur after the analysis. To round, consider the digit to the right of the last significant digit: if <5, then round down; if  $\geq 5$ , then round up. Means and medians will be presented with one more decimal place than the precision of the data. Standard deviations will be presented with two more decimal places than the precision of the data. Percentages will be presented with one decimal place. Minimums and maximums will be presented with the same precision as the original data.

All analyses will be performed using the SAS System® version 9.3 or higher. The domain (Study data tabulation Model [SDTM]) and analysis (Analysis Data Model [ADaM]) data sets will be taken as input to the SAS programs that generate the reportready tables, figures and listings. The submission ready SDTM and ADaM data sets will be provided to the sponsor along with display deliveries. The specifications for the domain data sets and analysis data sets will be provided in a separate document.

For all analyses, subjects will be analyzed by treatment group according to the actual product received during treatment, i.e., "as treated."

The following conventions will be used throughout the study analysis:

- Assessment visit times are defined by time of treatment administration.
- Baseline value is defined as the last valid measurement prior to the first treatment administration.

Date: 08Sep2017

Sponsor: Insys Development Co, Inc. Statistical Analysis Plan

Protocol Number: INS005-17-111

Change from baseline is defined as post-baseline value minus baseline value.

- Duration of an AE will be computed in days as the stop date of the event minus the start date plus 1. If reported as ongoing at the time of database lock, the stop date is defined as the date of the last visit or the last date of any AE for the subject in the database, whichever is later. Missing dates will be imputed as described in Section 7.2.
- The number of days in the study is computed as: Date of study completion /withdrawal - the date of first treatment administration (Day 1) + 1.
- If duplicate values are obtained at a given visit (e.g., repeated vital sign measurements), the last value will be used unless it is noted that the measurement was in error for that value. Values that compromise interpretation will not be used in summaries (e.g., values that were obtained post-dose will not be summarized as pre-dose values).

Sponsor: Insys Development Co, Inc.

Statistical Analysis Plan

Protocol Number: INS005-17-111 Date: 08Sep2017

#### 4. ANALYSIS POPULATIONS

#### 4.1 Efficacy Population

This study has no efficacy analysis and so no efficacy population.

#### 4.2 Safety Population

The safety population will include all subjects who received at least 1 dose of study drug.

#### 4.3 Disposition of Subjects

Subjects will be considered enrolled into the study only when they have received study drug. If a subject is randomized but does not receive study drug, they will not be counted in any summaries.

All enrolled subjects will be listed. Subjects who are screened and who fail screening or withdraw consent prior to randomization will not be entered into the database or presented in summaries or data listings. Subjects who are randomized, treated, subjects included in the safety population, subjects who complete follow-up as well as subjects who withdraw early from the study and the reason for withdrawal will be summarized by treatment group and overall in the subject disposition summary table.

#### 4.4 Major Protocol Deviations

Patient specific protocol deviation information will be collected on the CRF. Site specific deviations will be collected by the CRA and logged in the trip reports. will prepare a final Excel export of all CRF deviations and append to this Excel all Site specific deviations to create a final Excel Database of Deviations. All protocol deviations in this database will be designated as major or minor prior to CRF database lock by the sponsor's medical monitor. A major deviation is typically one that may affect the outcome, analysis or interpretation of the study. All protocol deviations will be presented in a by-subject listing.

#### 5. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

#### 5.1 Demographics and Baseline Characteristics

Demographic variables include age, gender, race, ethnicity, surgical procedure, and PONV risk factor. Baseline characteristics include height (cm), weight (kg), and BMI (kg/m2). Demographics and baseline characteristics will be presented in by-subject listings and summarized overall and by treatment group.

#### 5.2 Medical History

Medical history, as collected at screening, will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 19.0 and presented in a by-subject listing using the coded and verbatim history terms.

#### 5.3 Prior and Concomitant Medications/Surgeries Details

Prior medications/surgeries are those that stop prior to the start of the first study drug treatment administration. Any medication/therapy that stops at or after this time or with missing stop dates is considered concomitant medication/therapy.

Prior and concomitant medications are collected at screening and updated throughout the study as needed. Prior and concomitant medications will be coded using WHO/ATC classification index version March 2016 and summarized separately by drug class and preferred name, overall and by treatment group, for the safety population.

Prior and concomitant therapies will be presented in a by-subject listing of verbatim and coded terms. Non-medical therapies will appear in a separate data listing.

#### 6. MEASUREMENTS OF TREATMENT COMPLIANCE

#### 6.1 Study Medication Compliance

Sponsor: Insys Development Co, Inc.

The exposure to study medication during the treatment periods will be listed by-subject and summarized by descriptive statistics for both the inpatient and outpatient portions of the study, and overall. As the dose administration during the inpatient period is under the control of the study sites, compliance during that time will not be summarized.

Compliance of the subject during the outpatient portion of the study will be assessed by summarizing the number of doses taken during the outpatient portion of the trial, and by the average number of doses taken per day during the outpatient portion of the trial, calculated as the number of doses taken divided by the number of days the subject remains in the outpatient portion of the study.

Subjects assigned to standard of care during the outpatient portion of the trial were instructed to take study medication only when they experienced pain. Subjects assigned Buprenorphine were instructed to maintain the TID dosing for the entire outpatient period.

Sponsor: Insys Development Co, Inc.

Statistical Analysis Plan
Date: 08Sep2017

#### 7. SAFETY EVALUATION

Protocol Number: INS005-17-111

#### 7.1 Overview of Safety Analysis Methods

The primary safety endpoints are the incidence of TEAEs.

The secondary safety endpoints are as follows:

- Proportion of subjects using rescue medication for nausea
- Time to first use of rescue medication for nausea following each dose of the investigational product (IP)
- Total use of rescue medication for nausea over 0-8 hours, 0 to 24 hours, over 0 to 48 hours, over 0-72 hours and 0-7 days
- Pulse oximetry
- ECGs at 90 minutes, 12, 24, 48 and 72 hours
- Oral examinations

#### 7.2 Adverse Events

Treatment-emergent AEs are defined as AEs that start or worsen in severity after the first exposure to study medication. Verbatim terms used by investigators to identify AEs in the CRFs will be mapped to the appropriate preferred term (PT) and system organ class (SOC) using a standardized coding dictionary (MedDRA Version 19.0). All coding will be reviewed prior to database lock. All recorded AEs will be listed, but only TEAEs will be summarized.

A serious adverse event (SAE) is any AE that meets any of the following causes:

- Results in death;
- Is life-threatening;
- Requires in-subject hospitalization or prolongation of existing hospitalization;
- Results in persistent or significant disability or incapacity;
- Is a congenital anomaly or birth defect;
- Is medically significant or requires intervention to prevent one of the outcomes listed above.

Serious AEs will be captured from the time of consent through the end of the study.

An overall summary will be prepared giving, for each treatment group and overall, both the number of events, and the number of subjects with events for the following events:

Sponsor: Insys Development Co, Inc. CO

Protocol Number: INS005-17-111 Date: 08Sep2017

- all TEAEs.
- serious TEAEs
- treatment related TEAEs.
- SAEs and TEAEs leading to premature discontinuation of study.

In addition, the overall summary will be produced by the study stratification variables: PONV risk group and surgical procedure.

Incidence of TEAEs will be summarized for each treatment group by SOC and PT sorted in descending frequency by system organ class (SOC), and then by preferred term (PT) within SOC. Separate tables will be created for each of the following event sets:

- All TEAEs
- Treatment related TEAEs (defined as Possibly, Probably or Definitely related)
- TEAEs leading to premature discontinuation from study
- Serious AEs
- TEAEs by maximum severity

The following AE listings will be created: all AEs, treatment related AEs, serious AEs, deaths, and AEs leading to premature discontinuation.

If a given subject experiences a TEAE that maps to the same PT more than once, the subject will be counted once for the PT at its greatest severity (i.e., mild, moderate, or severe) and causality (i.e., attribution to treatment).

Duration of a TEAE will be computed in days as the stop date of the event minus the start date plus 1 and included in by subject listings. If reported as ongoing at the time of database lock, the stop date is defined as the date of the last visit or the last date of any event for the subject in the database, whichever is later. If a TEAE is considered resolved, but the stop date is missing, the last day of the month will be imputed if the month and year are available. If only the year is available, and the year is the same as the year of the last visit, the stop date will be the latest of the last visit date or latest event for the subject in the database. If the year of the event is prior to the year of the last treatment, the end day and month will be set to 31 December.

For missing or partial start dates, it is most conservative to impute them as temporally related to the first dose of study medication. The following chart will be used to impute start date:

Statistical Analysis Plan

Date: 08Sep2017

Sponsor: Insys Development Co, Inc.

Table 7-1 Table of AE Start Date Imputation Rules

Protocol Number: INS005-17-111

| | | Same as | |
|---|---|---|---|
| Missing Start | Prior to | Treatment Start | After Treatment Start |
| Date Portion | Treatment | Date | Date |
| Day | Month and Year < | Month and Year = | Month and Year > |
| | Month and Year of first | Month and Year of | Month and Year of |
| | treatment: | first treatment: | First Treatment: |
| | Day = 1 | Day = Day of first treatment | Day = 1 |
| Day and | Year < Year of first | Year = Year of | Year > Year of first |
| Month | treatment: | first treatment: | treatment: |
| | Day = 1, | Day = Day of first | Day = 1, |
| | Month = July | treatment, | Month = January |
| | | Month = Month of | • |
| | | first treatment | |
| Day, Month, | To be conservative, com | pletely missing start d | lates will be set to the |
| and Year | date of first treatment | _ | |

After following these imputation rules, if the start date is imputed as a date after the end date, the start date will be set to the end date to provide a positive duration for the event incidence.

Missing assessments for AE study medication relationship or severity will be summarized as definitely related or severe respectively. No other imputation is planned for safety data.

#### Rescue Medication 7.3

The total use of rescue and the proportion of patients given rescue medication for nausea relief will be summarized by treatment group and by cumulative time point (0-8 hours, 0-24 hours, 0-48 hours, 0-72 hours and 0-7 days) and overall. A by-subject listing presenting the use of nausea rescue medication over time will be given.

Time to first rescue medication for nausea is the time (in minutes) elapsed from the time of first dose of IP to time the first dose of rescue medication for nausea is given. A

summary table will present the median time to first rescue use and 95% confidence intervals of the medians by treatment group as determined by log-rank analysis performed using SAS PROC LIFETEST. A summary figure will present the time to first rescue use as a Kaplan-Meier survival plot. If a subject does not take rescue medication for nausea but prematurely discontinues from the study, then for analysis purposes the subject will be censored at the time of discontinuation. If a subject never takes rescue medication for nausea and completes the treatment phase of the study, then the subject will be considered censored for analysis purposes at 7 days.

#### 7.4 Clinical Laboratory Evaluation

The following clinical laboratory tests will be performed for individual subjects.

**Serum Chemistry**: Albumin, total bilirubin, total protein, calcium, alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, blood urea nitrogen, cholesterol, glucose, sodium, potassium, chloride, bicarbonate, lactate dehydrogenase, uric acid, creatinine with calculated creatinine clearance (Cockcroft-Gault method).

**Hematology**: Hemoglobin, hematocrit, red blood cell count, red blood cell indices, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, platelet count (or estimate), and white blood cell count including differential.

**Urinalysis**: pH, specific gravity, blood, glucose, protein, and ketones.

Baseline for clinical laboratory parameters will be defined as the last evaluation before dosing with study treatment. For each continuous parameter, summary statistics of values and change from baseline will be presented by treatment group and overall; categorical urinalysis test parameters will be summarized using number and proportion of normal and abnormal results at each visit. All clinical laboratory values will be listed.

#### 7.5 Vital Signs

Vital signs results including pulse oximetry, BP [systolic and diastolic], pulse rate, respiration rate, and body temperature will be listed for individual subjects. Baseline for vital signs measurements will be defined as the last evaluation before dosing with study medication. Summary statistics of values and changes from baseline to each study time point will be presented by treatment group and overall

#### 7.6 Physical, Oral and ECG Exams

All findings of physical, oral and ECG examinations will be listed for individual subjects and abnormal findings will be summarized by time point.

A physical exam will be conducted at screening, before surgery on Day 1, 72 hours (±4 hours) after first dose of study drug (Time 0), and at the Follow-up Visit/ET. Physical examination systems include HEENT, cardiovascular, respiratory, gastrointestinal, neurological, dermatologic, and musculoskeletal systems.

An oral cavity exam will consist of a sublingual assessment, noting the colour of mucosa and whether inflammation is present, a check for mucositis and local irritation. The oral cavity examinations should be conducted at screening, pre-surgery, before the first dose of study drug, and then at 90 minutes ( $\pm 10$  minutes), and at 12, 24, 48 hours, 72 hours ( $\pm 10$  minutes) after Time 0, and at Follow-up Visit/ET. Assessments will be repeated based on the Investigator's discretion.

The ECG will be evaluated for any clinically relevant cardiovascular conditions, defined as any clinically significant abnormalities identified by the reader related to coronary artery disease, coronary spasm, abnormal heart rhythm, hypertrophic cardiomyopathy, heart failure, rheumatic heart disease, or myocarditis. An ECG will be performed at screening, before the first dose of study drug, and then at 90 minutes ( $\pm 10$  minutes), and at 12, 24, 48 hours, 72 hours ( $\pm 10$  minutes) after Time 0 and at Follow-up Visit/ET

# 7.7 Serology Screens, Drug of Abuse and Alcohol Screens, Pregnancy Test

Results of, HIV and hepatitis B and C screens, drug of abuse and alcohol screens, and pregnancy tests will be listed for individual subjects. Each test result will be defined to be "negative" or "positive" according to the normal reference range from the clinical laboratory.

# 8. EFFICACY EVALUATION

There is to be no efficacy analysis in this study.

### 9. OTHER ANALYSES

Any additional analyses conducted will be considered exploratory and enumerated in the CSR.

### 10.INTERIM ANALYSES AND DATA MONITORING

There are no planned interim analyses for this study.

### 11. CHANGES TO THE ANALYSES PLANNED IN THE PROTOCOL

Any deviations from the statistical plan will be described and a justification given in the CSR.

Sponsor: Insys Development Co, Inc. CON

Protocol Number: INS005-17-111 Date: 08Sep2017

#### 12. REFERENCES

US Federal Register. (1998) *International Conference on Harmonization; Guidance for Industry: Statistical Principles for Clinical Trials*. Department of Health and Human Services: Food and Drug Administration. Federal Register, Vol. 63, No. 179, September 16, 1998, page 49583.

US Federal Register. (1996) *International Conference on Harmonization; Guidance for Industry: Structure and Content of Clinical Study Reports*. Department of Health and Human Services: Food and Drug Administration. Federal Register Vol. 61, July 17, 1996, page 37320.

Guidance for Industry (2014) *Analgesic Indications: Developing Drug and Biological Products - Draft Guidance*. Department of Health and Human Services: Food and Drug Administration. Center for Drug Evaluation and Research (CDER) February 2014 Clinical/Medical.

CONFIDENTIAL Statistical Analysis Plan

Protocol Number: INS005-17-111 Date: 08Sep2017

#### 13. APPENDICES

Sponsor: Insys Development Co, Inc.

# 13.1 List of Tables for Final Study Report

| Table 14.1.1 | All Subjects | Summary of Subject Disposition |
|---|---|---|
| Table 14.1.2 | Safety Population | Summary of Demographic and Baseline Characteristics |
| Table 14.1.3 | Safety Population | Summary of Prior Medications |
| Table 14.1.4 | Safety Population | Summary of Concomitant Medications |
| Table 14.1.5 | Safety Population | Summary of Study Medication Compliance (Outpatient) |
| Table 14.1.6 | Safety Population | Summary of Study Medication Exposure |
| Table 14.3.1.1.1 | Safety Population | Overall Summary of Treatment-Emergent Adverse Events (TEAEs) |
| Table 14.3.1.1.2 | Safety Population | Overall Summary of TEAEs By PONV Classification |
| Table 14.3.1.1.3 | Safety Population | Overall Summary of TEAEs By Type Of Surgery |
| Table 14.3.1.2 | Safety Population | Summary of TEAEs by System Organ Class (SOC) and Preferred Term (PT) |
| Table 14.3.1.3 | Safety Population | Summary of Treatment Related TEAEs by SOC and PT |
| Table 14.3.1.4 | Safety Population | Summary of SAEs by SOC and PT |

Sponsor: Insys Development Co, Inc. CONFIDENTIAL Statistical Analysis Plan

Protocol Number: INS005-17-111 Date: 08Sep2017

| Table 14.3.1.5 | Safety Population | Summary of TEAEs Leading To Study Drug Discontinuation by SOC and PT |
|---|---|---|
| Table 14.3.1.6 | Safety Population | Summary of TEAEs by System Organ Class, Preferred Term and Maximum Severity |
| Table 14.3.1.7 | Safety Population | Summary of Total Rescue Use and Proportion Of Subjects Using Rescue Medication For Nausea By Time Interval |
| Table 14.3.1.8 | Safety Population | Summary Of Time To First Rescue For Nausea |
| Table 14.3.2.1.1 | Safety Population | Summary of Chemistry Results by Study Visit |
| Table 14.3.2.1.2 | Safety Population | Summary of Hematology Results by Study Visit |
| Table 14.3.2.1.3 | Safety Population | Summary of Urinalysis Results by Study Visit Continuous Assays |
| Table 14.3.2.1.4 | Safety Population | Summary of Urinalysis Results by Study Visit Categorical Assays |
| Table 14.3.3 | Safety Population | Summary of Vital Signs and Changes from Baseline by Study Visit |
| Table 14.3.4 | Safety Population | Summary of Physical Exam Findings |
| Table 14.3.5 | Safety Population | Summary of Oral Cavity Exam Findings |
| Table 14.3.6 | Safety Population | Summary of ECG Exam Findings |
| Table 14.3.7 | Safety Population | Summary of ECG Results and Changes from Baseline by Study Visit |

Sponsor: Insys Development Co, Inc. CONFIDENTIAL Statistical Analysis Plan

Protocol Number: INS005-17-111 Date: 08Sep2017

# 13.2 List of Figures for Final Study Report

| Figure 14.1 | Safety Population | Time To First Use Of Rescue Medication for Nausea |
|---|---|---|

# 13.3 List of Listings for Final Study Report

| Listing 16.2.1.1 | All Subjects | Subject Enrollment and Randomization |
|---|---|---|
| Listing 16.2.1.3 | All Subjects | Subject Disposition |
| Listing 16.2.2.1 | Safety Population | Protocol Deviations |
| Listing 16.2.4.1 | Safety Population | Demographics and Baseline Characteristics |
| Listing 16.2.4.2 | Safety Population | Medical/Surgical History |
| Listing 16.2.4.3 | Safety Population | Prior and Concomitant Medications |
| Listing 16.2.4.4 | Safety Population | Non-Medication Therapy |
| Listing 16.2.4.5 | Safety Population | Serology Laboratory And Pregnancy Test Results |
| Listing 16.2.4.6 | Safety Population | Alcohol Breath Test And Urine Drug Screen |

| Sponsor: Insys Development Co, Inc | c. CONFIDENTIAL | Statistical Analysis Plan |
|---|---|---|
| Protocol Number: INS005-17-111 | | Date: 08Sep2017 |
| Listing 16.2.4.7 | Safety Population | Surgery |
| Listing 16.2.5.1 | Safety Population | Study Drug Administration |
| Listing 16.2.5.2 | Safety Population | Discharge To Outpatient Treatment |
| Listing 16.2.5.3 | Safety Population | Study Drug Accountability |
| Listing 16.2.5.4 | Safety Population | Rescue Medication Administration |
| Listing 16.2.7.1 | Safety Population | All Treatment Emergent Adverse Events (TEAEs) |
| Listing 16.2.7.2 | Safety Population | Treatment Related TEAEs |
| Listing 16.2.7.3 | Safety Population | Serious TEAEs |
| Listing 16.27.4 | Safety Population | Deaths |
| Listing 16.2.7.5 | Safety Population | TEAEs Leading To Study Drug Discontinuation |
| Listing 16.2.8.1.1 | Safety Population | Chemistry Laboratory Results |
| Listing 16.2.8.1.2 | Safety Population | Hematology Laboratory Results |
| Listing 16.2.8.1.3 | Safety Population | Urinalysis Laboratory Results |
| Listing 16.2.8.2 | Safety Population | Vital Signs |
| Listing 16.2.8.3.1 | Safety Population | Physical Examinations |
| Listing 16.2.8.3.2 | Safety Population | Oral Cavity Examinations |
| Sponsor: Insys Development Co, Inc | c. CONFIDENTIAL | Statistical Analysis Plan | |
|---|---|---|--|
| Protocol Number: INS005-17-111 | | Date: 08Sep2017 | |
| Listing 16.2.8.4 | Safety Population | ECG Exam Assessment | |
| Listing 16.2.8.5 | Safety Population | Comments | |

13.4 TABLE, FIGURE AND LISTING SPECIFICATIONS

Protocol No.: INS005-17-111 

| Table 14.1.1 Summary of Subject Disposition All Subjects |
|---|
| Table 14.1.2 Summary of Demographic and Baseline Characteristics Safety Population 43 |
| Table 14.1.3 Summary of Prior Medications [1] Safety Population 45 |
| Table 14.1.4 Summary of Concomitant Medications Safety Population 46 |
| Table 14.1.5 Summary of Study Medication Compliance (Outpatient) Safety Population 47 |
| Table 14.1.6 Summary of Study Medication Exposure Safety Population48 |
| Table 14.3.1.1.1 Overall Summary of Treatment-Emergent Adverse Events (TEAEs) Safety Population 49 |
| Table 14.3.1.1.2 Overall Summary of Treatment-Emergent Adverse Events (TEAEs) By PONV Classification Safety Population |
| Table 14.3.1.1.3 Overall Summary of Treatment-Emergent Adverse Events (TEAEs) By Type Of Surgery Safety Population |
| Table 14.3.1.2 Summary of TEAEs by System Organ Class (SOC) and Preferred Term (PT) Safety Population 55 |
| Table 14.3.1.3 Summary of Treatment Related TEAEs by SOC and PT Safety Population 56 |
| Table 14.3.1.4 Summary of SAEs by SOC and PT Safety Population 56 |
| Table 14.3.1.5 Summary of TEAEs Leading To Study Drug Discontinuation by SOC and PT Safety Population 56 |
| Table 14.3.1.6 Summary of TEAEs by System Organ Class, Preferred Term and Maximum Severity Safety Population57 |
| Table 14.3.1.7 Summary of Total Rescue Use and Proportion Of Subjects Using Rescue Medication For Nausea By Time Interval Safety Population58 |


| Table 14.3.1.8 Summary Of Time 10 First Rescue For Nausea Safety Population 59 | |
|---|---|
| Table 14.3.2.1.1 Summary of Chemistry Results by Study Visit Safety Population 60 | |
| Table 14.3.2.1.2 Summary of Hematology Results by Study Visit Safety Population 61 | |
| Table 14.3.2.1.3 Summary of Urinalysis Results by Study Visit Continuous Assays Safety Population | 61 |
| Table 14.3.2.1.4 Summary of Urinalysis Results by Study Visit Categorical Assays Safety Population | 62 |
| Table 14.3.3 Summary of Vital Signs and Changes From Baseline by Study Visit Safety Population | 63 |
| Table 14.3.4 Summary of Physical Exam Findings Safety Population 65 | |
| Table 14.3.5 Summary of Oral Cavity Exam Findings Safety Population . 66 | |
| Table 14.3.6 Summary of ECG Exam Findings Safety Population 67 | |
| Table 14.3.7 Summary of ECG Results and Changes from Baseline by Study Visit Safety Population | 68 |
| Figure 14.1 Time To First Use Of Rescue Medication Safety Population . 69 | |
| Listing 16.2.1.1 Subject Enrollment and Randomization All Subjects71 | |
| Listing 16.2.1.3 Subject Disposition All Subjects72 | |
| Listing 16.2.2.1 Protocol Deviations Safety Population | |
| Listing 16.2.4.1 Demographics and Baseline Characteristics Safety Population 74 | |
| Listing 16.2.4.2 Medical/Surgical History Safety Population | |
| Listing 16.2.4.3 Prior and Concomitant Medications Safety Population 76 | |
| Listing 16.2.4.4 Non-Medication Therapy Safety Population77 | |
| Listing 16.2.4.5 Serology Laboratory And Pregnancy Test Results Safety Population 78 | |

| Listing 16.2.4.6 Alcohol Breath Test and Urine Drug Screen[1] Safety | Population 79 | |
|---|---|---|
| Listing 16.2.4.7 Surgery Safety Population | 80 | |
| Listing 16.2.5.1 Study Drug Administration Safety Population | 81 | |
| Listing 16.2.5.2 Discharge to Outpatient Treatment Safety Population | 82 | |
| Listing 16.2.5.3 Study Drug Accountability Safety Population | 83 | |
| Listing 16.2.5.4 Rescue Medication Administration Safety Population | 84 | |
| Listing 16.2.7.1 All Treatment Emergent Adverse Events (TEAEs) Safe | ty Population | 85 |
| Listing 16.2.7.2 Treatment Related TEAEs Safety Population | 86 | |
| Listing 16.2.7.3 Serious TEAEs Safety Population | 86 | |
| Listing 16.2.7.4 Deaths Safety Population | 86 | |
| Listing 16.2.7.5 TEAEs Leading To Premature Study Discontinuation S | Safety Population | 86 |
| Listing 16.2.8.1.1 Chemistry Laboratory Results Safety Population | 87 | |
| Listing 16.2.8.1.2 Hematology Laboratory Results Safety Population | 88 | |
| Listing 16.2.8.1.3 Urinalysis Laboratory Results Safety Population | 89 | |
| Listing 16.2.8.2 Vital Signs Safety Population | 90 | |
| Listing 16.2.8.3.1 Physical Examinations Safety Population | 91 | |
| Listing 16.2.8.3.2 Oral Cavity Examinations Safety Population | 92 | |
| Listing 16.2.8.4 ECG Exam Assessment Safety Population | 93 | |
| Listing 16.2.8.5 Comments Safety Population | 94 | |


Sponsor: Insys Development Company, Inc

# 14. GENERAL PROGRAMMING NOTES

All continuous study assessments will be summarized by treatment and time point (as applicable) using descriptive statistics (n, mean, standard deviation, median, and range (minimum, maximum)). All categorical study assessments will be summarized by treatment and time point (as applicable) using frequency counts and percentages. All study data will be listed by treatment group, subject and time point (as applicable).

No preliminary rounding should be performed; rounding should only occur after analysis. To round, consider digit to right of last significant digit: if < 5 then round down, if  $\ge 5$  then round up. Means and medians will be presented with one more decimal place than the precision of the data. Standard deviations will be presented with two more decimal places than the precision of the data. Percentages will be presented with one decimal place. Minimums and maximums will be presented with the same precision as the original data.

# **Study Conventions:**

- Day 1 is the day of baseline and first exposure study treatment.
- Assessment time point times are defined by time after administration of study drug.
- Baseline value is defined as the last valid measurement prior to treatment.
- Change from baseline is defined as post-baseline value minus baseline value.
- Duration of an adverse event will be computed in days as the [stop date of the event minus the start date] plus 1. See SAP for imputation rules for missing dates.
- The number of days in the study is computed as: [Date of study completion (or withdrawal) the date of first dose (Day 1)] + 1.
- If duplicate values are obtained at a given time point (e.g., repeated vital sign measurements), the last value will be used unless it is noted that the measurement was in error for that value. Values that compromise interpretation will not be used in summaries (e.g., values that were obtained post-dose will not be summarized as pre-dose values).


Sponsor: Insys Development Company, Inc

Table 14.1.1
Summary of Subject Disposition
All Subjects

| | Standard Narcotic Therapy[1] N=xxx | Buprenorphine SL<br>Spray (0.5 mg TID)<br>N=xxx | Overall<br>N=xxx |
|---|---|---|---|
| Subjects Randomized | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Subjects in Safety Population (received treatment), n (%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Subjects completing study, n (%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Completed Inpatient Treatment/Completed Outpatient Treatment/Completed Follow-up | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Completed Inpatient Treatment/ Not Completed Outpatient Treatment/ Not Completed Follow-up | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Completed Inpatient Treatment/Completed Outpatient Treatment/ Not Completed Follow-up | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Treatment/Not completed Outpatient Treatment/ Not completed Follow-up | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| • | | | |
| Subjects with early termination, n (%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Adverse event, n (%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Death, n (%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Withdrawal of consent by subject, n (%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Subject Non-compliance, n (%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Protocol Violation, n (%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Lost to follow-up, n (%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Other, n (%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |

# Footnote:

[1] Subjects assigned Standard Narcotic Therapy were given morphine IV 4 mg TID for 24 hours, followed by Oxycodone Hydrochloride tablet, 10 mg TID for the remainder of the treatment period.


Table 14.1.2
Summary of Demographic and Baseline Characteristics
Safety Population

| | Standard Narcotic Therapy[1] | Buprenorphine SL Spray (0.5 mg TID) | Overall |
|---|---|---|---|
| | N = xx | N = xx | N = xx |
| Age | | | |
| N | XXX | XXX | XXX |
| Mean (SD) | XXX.X (XX.X) | XXX.X (XX.X) | XXX.X (XX.X) |
| Median | XXX | XXX | XXX |
| Range (Min, Max) | XXX, XXX | XXX, XXX | XXX, XXX |
| Sex, n (%) | | | |
| Male | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Female | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Race, n (%) | | | |
| White | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Black or African American | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Asian | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| American Indian or Alaskan Native | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Native Hawaiian or Pacific Islander | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Multiple | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Other | | | |
| Ethnicity, n (%) | | | |
| Hispanic or Latino | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Non-Hispanic or Latino | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Unknown | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Baseline Height (cm) | | | |
| N | XXX | XXX | XXX |
| Mean (SD) | XXX.X (XX.X) | XXX.X (XX.X) | XXX.X (XX.X) |
| Median | XXX | XXX | XXX |
| Range (Min, Max) | XXX, XXX | XXX, XXX | XXX, XXX |


Sponsor: Insys Development Company, Inc

| | Standard Narcotic Therapy[1] | Buprenorphine SL Spray (0.5 mg TID) | Overall |
|---|---|---|---|
| | N = xx | N = xx | N = xx |
| Baseline Weight (kg) | | | |
| N | XXX | XXX | XXX |
| Mean (SD) | XXX.X (XX.X) | XXX.X (XX.X) | XXX.X (XX.X) |
| Median | XXX | XXX | XXX |
| Range (Min, Max) | XXX, XXX | XXX, XXX | XXX, XXX |
| Baseline BMI (kg/m²) [2] | | | |
| N | XXX | XXX | XXX |
| Mean (SD) | XXX.X (XX.X) | XXX.X (XX.X) | XXX.X (XX.X) |
| Median | XXX | XXX | XXX |
| Range (Min, Max) | XXX, XXX | XXX, XXX | XXX, XXX |
| Baseline PONV Risk Factor | | | |
| 0 | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| 1 | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| 2 | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| 3 | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| 4 | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Baseline PONV Risk Factor | | | |
| Low Risk | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| High Risk | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Surgical Procedure | | | |
| Bunionectomy | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Breast Implant | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Abdominoplasty | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |

#### Footnotes:

Percentages are based on the number of subjects (N) in a given treatment group for the population analyzed.

# Programmer Notes:

For categorical variables, missing categories (e.g. no Hispanics) should appear with an n and % of zero.

<sup>[1]</sup> Subjects assigned Standard Narcotic Therapy were given morphine IV 4 mg TID for 24 hours, followed by Oxycodone Hydrochloride tablet, 10 mg TID for the remainder of the treatment period.

<sup>[2]</sup> BMI is calculated as BMI = Weight(kg) / [Height(m)^2].


Sponsor: Insys Development Company, Inc

Table 14.1.3
Summary of Prior Medications [1]
Safety Population

| System Organ Class<br>Preferred Term | Standard Narcotic Buprenorphine SL Spray (0.5 Therapy[2] mg TID) | | Overall |
|---|---|---|---|
| | N=xx | N=xx | N=xx |
| Number of Subjects with Any Prior Medication, | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| n (%) [3] | | | |
| ATC Class 1[4] | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Preferred Term 1 | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Preferred Term 2 | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| ATC Class 2 | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Preferred Term 1 | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Preferred Term 2 | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Etc. | | | |

#### Footnotes:

- [1] Prior medications include all medications that were started and stopped prior to study drug initiation.
- [2] Subjects assigned Standard Narcotic Therapy were given morphine IV 4 mg TID for 24 hours, followed by Oxycodone Hydrochloride tablet, 10 mg TID for the remainder of the treatment period.
- [3] n = Number of subjects reporting at least one medication within an ATC Class and Preferred Term; (%) = Percentage of subjects among Treatment Group (N). A subject reporting more than one medication for a particular ATC Class or Preferred Term is counted only once for each ATC Class or Preferred Term.
- [4] ATC Class and Preferred Term are based on the WHO/ATC classification index version March 2016 drug coding dictionary.

#### Programmer Notes:

Table entries should be sorted in decreasing order by overall n of ATC Class and by PT overall n within ATC Class based on the pooled EB-001 column.


Sponsor: Insys Development Company, Inc

Table 14.1.4
Summary of Concomitant Medications
Safety Population

| System Organ Class Preferred Term | Standard Narcotic Therapy[1] | Buprenorphine SL Spray (0.5 mg TID) |
|---|---|---|
| | N=xx | N=xx |
| Number of Subjects with Any Concomitant Medication, n (%) | XXX (XX.X%) | XXX (XX.X%) |
| ATC Class 1 Preferred Term 1 | XXX (XX.X%)<br>XXX (XX.X%) | XXX (XX.X%) XXX (XX.X%) |
| Preferred Term 2 | XXX (XX.X%) | XXX (XX.X%) |
| ATC Class 2 | XXX (XX.X%) | XXX (XX.X%) |
| Preferred Term 1 | XXX (XX.X%) | XXX (XX.X%) |
| Preferred Term 2 Etc. | XXX (XX.X%) | XXX (XX.X%) |

#### Footnotes:

- [1]Concomitant medications include all medications that were started or stopped after study drug initiation or those with missing stop dates.
- [2] Subjects assigned Standard Narcotic Therapy were given morphine IV 4 mg TID for 24 hours, followed by Oxycodone Hydrochloride tablet, 10 mg TID for the remainder of the treatment period.
- [3] n = Number of subjects reporting at least one medication within an ATC Class and Preferred Term; (%) = Percentage of subjects among Treatment Group (N). A subject reporting more than one medication for a particular ATC Class or Preferred Term is counted only once for each ATC Class or Preferred Term.
- [4] ATC Class and Preferred Term are based on the WHO/ATC classification index version March 2016 drug coding dictionary.

# Programmer Notes:

Table entries should be sorted in decreasing order by overall n of ATC Class and by PT n within ATC Class based on the pooled EB-001 column.


Sponsor: Insys Development Company, Inc

Table 14.1.5
Summary of Study Medication Compliance (Outpatient)
Safety Population

| | Standard Narcotic | Buprenorphine SL Spray | Overall |
|---|---|---|---|
| | Therapy[1] | (0.5 mg TID) | |
| | N = xx | N = xx | N = xx |
| Total Number of Doses taken during Outpatient period | | | |
| [2] | | | |
| n | X | X | X |
| Mean | X.X | X.X | X.X |
| SD | X.XX | X.XX | X.XX |
| Median | X.X | X.X | X.X |
| Range (Min, Max) | (X.X - X.X) | (X.X - X.X) | (X.X - X.X) |
| Average Number of Doses per Day During Outpatient | | | |
| Average Number of Doses per Day During Outpatient period [3] | | | |
| | x | Х | X |
| period [3] | x<br>x.x | х<br>х.х | х<br>х.х |
| period [3] | | | |
| period [3] n Mean | X.X | X.X | X.X |

#### Footnote:

- [1] Subjects assigned Standard Narcotic Therapy were given morphine IV 4 mg TID for 24 hours, followed by Oxycodone Hydrochloride tablet, 10 mg TID for the remainder of the treatment period.
- [2] The number of doses taken is the number dispensed number returned. Subjects assigned Standard Narcotic Therapy during the outpatient portion of the trial were instructed to take study medication only when they experienced pain. Subjects assigned Buprenorphine SL Spray (0.5 mg TID) were instructed to maintain the TID dosing for the entire outpatient period.
- [3] Average number of doses is calculated as the number of doses taken divided by the number of days the subject remained in the outpatient portion of the study.


Sponsor: Insys Development Company, Inc

Table 14.1.6
Summary of Study Medication Exposure
Safety Population

| | Standard Narcotic Therapy [1] | | Buprenorphine SL Spray<br>(0.5 mg TID) [2] |
|---|---|---|---|
| | Morphine | Oxycodone | |
| | N = xx | N = xx | N = xx |
| Total Exposure during Inpatient period (mg) | | | |
| n | X | X | X |
| Mean | X.X | X.X | X.X |
| SD | X.XX | X.XX | X.XX |
| Median | X.X | X.X | X.X |
| Range (Min, Max) | (X.X - X.X) | (X.X - X.X) | (X.X - X.X) |
| Total Exposure during Outpatient period (mg) [3] | | | |
| n | | X | X |
| Mean | | X.X | X.X |
| SD | | X.XX | X.XX |
| Median | | X.X | X.X |
| Range (Min, Max) | | (X.X - X.X) | (X.X - X.X) |
| Total Exposure Overall (mg) | | | |
| n | X | X | X |
| Mean | X.X | X.X | X.X |
| SD | X.XX | X.XX | X.XX |
| Median | X.X | X.X | X.X |
| Range (Min, Max) | (X.X - X.X) | (X.X - X.X) | (X.X - X.X) |

## Footnotes:

<sup>[1]</sup> Subjects assigned Standard Narcotic Therapy were given morphine IV 4 mg TID for 24 hours, followed by Oxycodone Hydrochloride tablet, 10 mg TID for the remainder of the treatment period.

<sup>[2]</sup> Subjects assigned to Buprenorphine SL Spray (0.5 mg TID) received Buprenorphine sublingual spray 0.5 mg TID for the entire treatment period.

<sup>[3]</sup> During the outpatient portion of the trial, subjects assigned to Standard Narcotic Therapy were instructed to take study medication only when they experienced pain, while subjects assigned to Buprenorphine SL Spray (0.5 mg TID) were instructed to maintain the TID dosing for the entire outpatient period.


Sponsor: Insys Development Company, Inc

Table 14.3.1.1.1

Overall Summary of Treatment-Emergent Adverse Events (TEAEs)

Safety Population

| | Standard Narcotic Therapy[4] | Buprenorphine SL<br>Spray (0.5 mg TID) | Overall |
|---|---|---|---|
| | N=xx | N=xx | N=xx |
| Number of TEAEs Reported | XX | XX | XX |
| Number of Subjects with Any TEAEs Reported [1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Number of Treatment related TEAEs Reported | XX | XX | XX |
| Number of Subjects with Treatment related TEAE Reported [1][2] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Number of Serious TEAEs Reported | | | |
| Number of Subjects with Any Serious TEAE Reported [1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Number of Subjects with TEAEs by Severity [3] | | | |
| Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Severe | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Number of Subjects with TEAEs Resulting in Study Drug<br>Discontinuation | | | |

#### Footnotes:

- [1] Subjects are only counted once at each level of summarization.
- [2] AEs are considered treatment related if they are identified as definitely, probably or possibly treatment (study drug) related. They are considered unrelated if they are identified as unlikely related or not related.
- [3] Subjects are counted once under the maximum severity if a subject experiences multiple adverse events.
- AEs with 'Severity Unknown or Not Reported' are summarized as serious AEs in summary tables by system organ class and preferred term.
- [4] Subjects assigned Standard Narcotic Therapy were given morphine IV 4 mg TID for 24 hours, followed by Oxycodone Hydrochloride tablet, 10 mg TID for the remainder of the treatment period.

Programming Note: The row 'Number of AEs Reported' displays the number of unique AE counts. For example, if a subject has the same AE (same preferred term) more than once, the subject is counted only once for the same AE. If a subject has different AEs (like headache


Sponsor: Insys Development Company, Inc

and skin rash), then the subject is counted more than once. (In other words, a subject is counted more than once for different AEs, but only once for the same AE occurring multiple times).


Sponsor: Insys Development Company, Inc

Table 14.3.1.1.2

Overall Summary of Treatment-Emergent Adverse Events (TEAEs) By PONV Classification Safety Population

| PONV | | Low Risk | | | High Risk | |
|---|---|---|---|---|---|---|
| | Standard<br>Narcotic<br>Therapy[4] | Buprenorphine<br>SL Spray (0.5<br>mg TID) | Overall | Standard<br>Narcotic<br>Therapy[4] | Buprenorphine<br>SL Spray (0.5<br>mg TID) | Overall |
| | N=xx | N=xx | N=xx | N=xx | N=xx | N=xx |
| Number of TEAEs Reported | XX | XX | XX | XX | XX | XX |
| Number of Subjects with Any TEAEs Reported [1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Number of Treatment related TEAEs Reported | XX | XX | XX | XX | XX | XX |
| Number of Subjects with Treatment related TEAE Reported [1][2] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Number of Serious TEAEs Reported<br>Number of Subjects with Any Serious TEAE<br>Reported [1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Number of Subjects with TEAEs by Severity [3] | | | | | | |
| Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Severe | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Number of Subjects with TEAEs Resulting in Study Drug Discontinuation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

#### Footnotes:

- [1] Subjects are only counted once at each level of summarization.
- [2] AEs are considered treatment related if they are identified as definitely, probably or possibly treatment related. They are considered unrelated if they are identified as unlikely related or not related.
- [3] Subjects are counted once under the maximum severity if a subject experiences multiple adverse events.
- AEs with 'Severity Unknown or Not Reported' are summarized as serious AEs in summary tables by system organ class and preferred term.
- [4] Subjects assigned Standard Narcotic Therapy were given morphine IV 4 mg TID for 24 hours, followed by Oxycodone Hydrochloride tablet, 10 mg TID for the remainder of the treatment period.


Sponsor: Insys Development Company, Inc

Programming Note: The row 'Number of AEs Reported' displays the number of unique AE counts. For example, if a subject has the same AE (same preferred term) more than once, the subject is counted only once for the same AE. If a subject has different AEs (like headache and skin rash), then the subject is counted more than once. (In other words, a subject is counted more than once for different AEs, but only once for the same AE occurring multiple times).


Table 14.3.1.1.3

Overall Summary of Treatment-Emergent Adverse Events (TEAEs) By Type Of Surgery Safety Population

| Surgery Type | | Bunionectomy | | Bre | ast Augmentat | | | Abdominoplast | Y |
|---|---|---|---|---|---|---|---|---|---|
| | Standard<br>Narcotic<br>Therapy[4] | Buprenor-<br>phine SL<br>Spray (0.5<br>mg TID) | Overall | Standard<br>Narcotic<br>Therapy[4] | Buprenor-<br>phine SL<br>Spray (0.5<br>mg TID) | Overall | Standard<br>Narcotic<br>Therapy[4] | Buprenor-<br>phine SL<br>Spray (0.5<br>mg TID) | Overall |
| | N=xx | N=xx | N=xx | N=xx | N=xx | N=xx | N=xx | N=xx | N=xx |
| Number of TEAEs<br>Reported | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Number of Subjects<br>with Any TEAEs<br>Reported [1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Number of<br>Treatment<br>related TEAEs<br>Reported [2] | xx | XX | XX | XX | XX | XX | XX | XX | XX |
| Number of Subjects<br>with Treatment<br>related TEAE<br>Reported [1][2] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Number of Serious<br>TEAEs Reported<br>Number of Subjects<br>with Any<br>Serious TEAE<br>Reported [1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Number of Subjects with TEAEs by Severity [3] Mild Moderate Severe | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) |


Sponsor: Insys Development Company, Inc

| Surgery Type | | Bunionectomy | | Bre | ast Augmentat | ion | 1 | Abdominoplasty | ? |
|---|---|---|---|---|---|---|---|---|---|
| | Standard<br>Narcotic<br>Therapy[4] | Buprenor-<br>phine SL<br>Spray (0.5<br>mg TID) | Overall | Standard<br>Narcotic<br>Therapy[4] | Buprenor-<br>phine SL<br>Spray (0.5<br>mg TID) | Overall | Standard<br>Narcotic<br>Therapy[4] | Buprenor-<br>phine SL<br>Spray (0.5<br>mg TID) | Overall |
| | N=xx | N=xx | N=xx | N=xx | N=xx | N=xx | N=xx | N=xx | N=xx |
| Number of Subjects with TEAEs Resulting in Study Drug Discontinuation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

#### Footnotes:

- [1] Subjects are only counted once at each level of summarization.
- [2] AEs are considered treatment related if they are identified as definitely, probably or possibly treatment related. They are considered unrelated if they are identified as unlikely related or not related.
- [3] Subjects are counted once under the maximum severity if a subject experiences multiple adverse events.
- AEs with 'Severity Unknown or Not Reported' are summarized as serious AEs in summary tables by system organ class and preferred term.
- [4] Subjects assigned Standard Narcotic Therapy were given morphine IV 4 mg TID for 24 hours, followed by Oxycodone Hydrochloride tablet, 10 mg TID for the remainder of the treatment period.

Programming Note: The row 'Number of AEs Reported' displays the number of unique AE counts. For example, if a subject has the same AE (same preferred term) more than once, the subject is counted only once for the same AE. If a subject has different AEs (like headache and skin rash), then the subject is counted more than once. (In other words, a subject is counted more than once for different AEs, but only once for the same AE occurring multiple times).


Sponsor: Insys Development Company, Inc

| System Organ Class Preferred Term | Standard Narcotic<br>Therapy[1]<br>N=xx | Buprenorphine SL Spray (0.5 mg TID) N=xx | Overall<br>N=xx |
|---|---|---|---|
| | n (%) #AEs | n (%) #AEs | n (%) #AEs |
| Subjects with any TEAE [Overall Number of AEs] | XX (XX.X%) [XX] | XX (XX.X%) [XX] | XX (XX.X%) [XX] |
| System Organ Class 1 | XX (XX.X%) [XX] | XX (XX.X%) [XX] | XX (XX.X%) [XX] |
| Preferred Term 1 | XX (XX.X%) [XX] | XX (XX.X%) [XX] | XX (XX.X%) [XX] |
| Preferred Term 2 | XX (XX.X%) [XX] | XX (XX.X%) [XX] | XX (XX.X%) [XX] |
| System Organ Class 2 | XX (XX.X%) [XX] | XX (XX.X%) [XX] | XX (XX.X%) [XX] |
| Preferred Term 1 | XX (XX.X%) [XX] | XX (XX.X%) [XX] | XX (XX.X%) [XX] |
| Preferred Term 2 | XX (XX.X%) [XX] | XX (XX.X%) [XX] | XX (XX.X%) [XX] |

#### Footnotes:

[1] Subjects assigned Standard Narcotic Therapy were given morphine IV 4 mg TID for 24 hours, followed by Oxycodone Hydrochloride tablet, 10 mg TID for the remainder of the treatment period.

Subjects are counted only once at each level of summarization (SOC or PT).

Summaries are sorted by SOC and PT within SOC by descending order of frequency of subjects.

 $\hbox{System Organ Class and Preferred Term are based on the Version 19.0 of the $MedDRA$ coding dictionary. } \\$ 

# Programmer Notes:

Table entries should be sorted in decreasing order by overall n of SOC and then by PT n within SOC based on the pooled EB-001 column.


Sponsor: Insys Development Company, Inc

Non-unique tables:

Table 14.3.1.3

Summary of Treatment Related TEAEs by SOC and PT
Safety Population

#### Programmer Notes:

- 1) Change row label 'Subjects With Any TEAE' to 'Subjects With Any Treatment Related TEAE'
- 2) Table entries should be sorted in decreasing order by overall n of SOC and then by PT n within SOC based on the pooled EB-001 column

Table 14.3.1.4
Summary of SAEs by SOC and PT
Safety Population

## Programmer Notes:

- 1) Change row label 'Subjects With Any TEAE' to 'Subjects With Any SAE'
- 2) Table entries should be sorted in decreasing order by overall n of SOC and then by PT n within SOC based on the pooled EB-001 column.

Table 14.3.1.5

Summary of TEAEs Leading To Study Drug Discontinuation by SOC and PT

Safety Population

# Programmer Notes:

- 1) Change row label 'Subjects With Any TEAE' to 'Subjects With Any TEAE Leading to Discontinuation'
- 2) Table entries should be sorted in decreasing order by overall n of SOC and then by PT n within SOC based on the pooled EB-001 column.


Sponsor: Insys Development Company, Inc

Table 14.3.1.6

Summary of TEAEs by System Organ Class, Preferred Term and Maximum Severity Safety Population

| | Standard | d Narcotic Th | erapy[1] | Buprenorp | phine SL Spra | y (0.5 mg | | Overall | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | TID) | | | | |
| | | N = xx | | | N = xx | | | N = xx | |
| | Mild | Moderate | Severe | Mild | Moderate | Severe | Mild | Moderate | Severe |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Patients with any TEAE | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| System Organ Class 1 | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Preferred Term 1 | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Preferred Term 2 | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Etc. | | | | | | | | | |

#### Footnotes:

[1] Subjects assigned Standard Narcotic Therapy were given morphine IV 4 mg TID for 24 hours, followed by Oxycodone Hydrochloride tablet, 10 mg TID for the remainder of the treatment period.

Subjects are counted only once at each level of summarization (SOC or PT). A patient will be counted once in each row of the table at the maximum severity reported for that system organ class or preferred term.

Patients missing severity for an AE are categorized as severe for that AE.

## Programmer Notes:

Table entries should be sorted in decreasing order by overall n of SOC and then by PT n within SOC based on the pooled EB-001 column.


Sponsor: Insys Development Company, Inc

Table 14.3.1.7

Summary of Total Rescue Use and Proportion Of Subjects Using Rescue Medication For Nausea By Time Interval Safety Population

| | Standard Narcotic Therapy[1] | Buprenorphine SL Spray (0.5 mg | Overall |
|---|---|---|---|
| | | TID) | |
| | N=xx | N=xx | N=xx |
| Total Use of Rescue for Nausea | | | |
| (number of doses) | | | |
| Within 0-8 Hours | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Within 0-24 Hours | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Within 0-48 Hours | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Within 0-72 Hours | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Within 0-7 Days | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| At any time during the | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| treatment period | | | |
| Proportion of Subjects given | | | |
| Rescue for Nausea | | | |
| Within 0-8 Hours | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Within 0-24 Hours | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Within 0-48 Hours | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Within 0-72 Hours | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Within 0-7 Days | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| At any time during the treatment period | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

## Footnote:

[1] Subjects assigned Standard Narcotic Therapy were given morphine IV 4 mg TID for 24 hours, followed by Oxycodone Hydrochloride tablet, 10 mg TID for the remainder of the treatment period.


Sponsor: Insys Development Company, Inc

Table 14.3.1.8

Summary Of Time To First Rescue For Nausea

Safety Population

| | Standard Narcotic Therapy[4] (N = XX) | Buprenorphine SL Spray (0.5 mg TID) (N = XX) | Overall (N = XX) |
|---|---|---|---|
| Time to First Rescue use for Nausea (min) | | | |
| Median Time [1] Range (Min,max) [2] | XXX | XXX | XXX |
| 95% CI [3] | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) |
| Censored Observations n (%)[4] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects receiving nausea rescue medication n (%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

## Footnotes:

- [1] Median Time = Median time to first use of nausea rescue medication.
- [2] Min and Max of uncensored observations.
- [3] CI = Confidence Interval.
- [4] If a subject does not take rescue medication for nausea but prematurely discontinues from the study, then the subject will be censored at the time of discontinuation. If a subject never takes rescue medication for nausea and completes the treatment phase of the study, then the subject will be considered censored at 7 days.
- [5] Subjects assigned Standard Narcotic Therapy were given morphine IV 4 mg TID for 24 hours, followed by Oxycodone Hydrochloride tablet, 10 mg TID for the remainder of the treatment period.


Sponsor: Insys Development Company, Inc

Table 14.3.2.1.1 Summary of Chemistry Results by Study Visit Safety Population

| | | | Albumen (for example | e) | | |
|---|---|---|---|---|---|---|
| | Standard Narcotic Therapy[1] N=XX | | | Buprenorphine SL Spray (0.5 mg TID) N=xx | | rall<br>=xx |
| Time point<br>Statistic | Value | Change From<br>Baseline | Value | Change From<br>Baseline | Value | Change From<br>Baseline |
| Screening (Baseline) N Mean (SD) Median Range (Min, Max) | XXX<br>XX.X (XX.XX)<br>XXX<br>(XXX, XXX) | | XXX<br>XX.X (XX.XX)<br>XXX<br>(XXX, XXX) | | XXX<br>XX.X (XX.XX)<br>XXX<br>(XXX, XXX) | |
| Follow-up N Mean (SD) Median Range (Min, Max) | XXX<br>XX.X (XX.XX)<br>XXX<br>(XXX, XXX) | XXX<br>XX.X (XX.XX)<br>XXX<br>(XXX, XXX) | XXX<br>XX.X (XX.XX)<br>XXX<br>(XXX, XXX) | XXX<br>XX.X (XX.XX)<br>XXX<br>(XXX, XXX) | XXX<br>XX.X (XX.XX)<br>XXX<br>(XXX, XXX) | XXX<br>XX.X (XX.XX)<br>XXX<br>(XXX, XXX) |

# Footnote:

[1] Subjects assigned Standard Narcotic Therapy were given morphine IV 4 mg TID for 24 hours, followed by Oxycodone Hydrochloride tablet, 10 mg TID for the remainder of the treatment period.

# Programmer note:

Chemistry parameters are listed alphabetically.

Include scheduled time points only.

Include the following for Serum Chemistry: albumin, total bilirubin, total protein, calcium, alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, blood urea nitrogen, cholesterol, glucose, sodium, potassium, chloride, bicarbonate, lactate dehydrogenase, uric acid, creatinine with calculated creatinine clearance (Cockcroft-Gault method).


Sponsor: Insys Development Company, Inc

Non-unique tables:

# Table 14.3.2.1.2 Summary of Hematology Results by Study Visit Safety Population

#### Footnotes:

[1] Subjects assigned Standard Narcotic Therapy were given morphine IV 4 mg TID for 24 hours, followed by Oxycodone Hydrochloride tablet, 10 mg TID for the remainder of the treatment period.

#### Programmer note:

Hematology parameters are listed alphabetically.

Include scheduled time points only.

Include the following for hematology values: Hemoglobin, hematocrit, red blood cell count, red blood cell indices, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, platelet count (or estimate), and white blood cell count including differential.

Table 14.3.2.1.3

Summary of Urinalysis Results by Study Visit

Continuous Assays

Safety Population

#### Footnotes:

[1] Subjects assigned Standard Narcotic Therapy were given morphine IV 4 mg TID for 24 hours, followed by Oxycodone Hydrochloride tablet, 10 mg TID for the remainder of the treatment period.

## Programmer note:

Laboratory parameters are listed alphabetically

Include scheduled time points only.

Include continuous urinalysis assays only.


Sponsor: Insys Development Company, Inc

Table 14.3.2.1.4

Summary of Urinalysis Results by Study Visit

Categorical Assays

Safety Population

| pH (for example) | | | |
|---|---|---|---|
| System Organ Class Preferred Term | Standard Narcotic | Buprenorphine SL Spray (0.5 | Overall |
| | Therapy[1] | mg TID) | |
| | N=xx | N=xx | N=xx |
| Lab Parameter | | | |
| Screening (Baseline) | | | |
| Category 1 | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Category 2 | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Category 3 | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Category 4 | XXX (XX.X%) | | |
| | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Follow-up | | | |
| Category 1 | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Category 2 | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Category 3 | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Category 4 | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |

Footnote:

Footnotes:

[1] Subjects assigned Standard Narcotic Therapy were given morphine IV 4 mg TID for 24 hours, followed by Oxycodone Hydrochloride tablet, 10 mg TID for the remainder of the treatment period.

Programmer note:

Laboratory parameters are listed alphabetically

Include scheduled time points only.

Include categorical urinalysis assays only.


Sponsor: Insys Development Company, Inc

Table 14.3.3

Summary of Vital Signs and Changes From Baseline by Study Visit
Safety Population

| | | Systolic blood pre | ssure (mmHg) (for | example) | | |
|---|---|---|---|---|---|---|
| | | tic Therapy[2]<br>XX | Buprenorphine SL Spray (0.5 mg<br>TID)<br>N=XX | | | rall<br>=XX |
| Study Visit/ Time point [1] Statistic | Actual | Change From<br>Baseline | Actual | Change From<br>Baseline | Actual | Change From<br>Baseline |
| Screening (Baseline) | | | | | • | • |
| n<br>Mean (S.D.)<br>Median<br>Range (Min, Max) | XXX<br>XX.X (XX.XX)<br>XXX<br>(XXX, XXX) | | XXX<br>XX.X (XX.XX)<br>XXX<br>(XXX, XXX) | | XXX<br>XX.X (XX.XX)<br>XXX<br>(XXX, XXX) | |
| Pre-surgery | | | | | | |
| n | XXX | XXX | XXX | XXX | XXX | XXX |
| Mean (S.D.))<br>Median<br>Range (Min, Max) | XX.X (XX.XX) XXX (XXX, XXX) | XX.X (XX.XX) XXX (XXX, XXX) | XX.X (XX.XX) XXX (XXX, XXX) | XX.X (XX.XX) XXX (XXX, XXX) | XX.X (XX.XX) XXX (XXX, XXX) | XX.X (XX.XX) XXX (XXX, XXX) |
| Pre-dose | | | | | | |
| n | XXX | XXX | XXX | XXX | XXX | XXX |
| Mean (S.D.))<br>Median<br>Range (Min, Max) | XX.X (XX.XX) XXX (XXX, XXX) | XX.X (XX.XX) XXX (XXX, XXX) | XX.X (XX.XX) XXX (XXX, XXX) | XX.X (XX.XX) XXX (XXX, XXX) | XX.X (XX.XX) XXX (XXX, XXX) | XX.X (XX.XX) XXX (XXX, XXX) |
| Etc. | | | | | | |

## Footnotes:

# [1] During treatment period:

Blood Pressure will be measured every 4 hours after first dose.

Pulse rate and respiratory rate will be measured at TO, 1h and every 2 hours after first dose.

Pulse Oximetry will be measured at 90 min, 12h, 24h, 48h, and 72h after first dose.

[2] Subjects assigned Standard Narcotic Therapy were given morphine IV 4 mg TID for 24 hours, followed by Oxycodone Hydrochloride tablet, 10 mg TID for the remainder of the treatment period.


Sponsor: Insys Development Company, Inc

Programmer note: Vital signs are: Systolic and diastolic blood pressure, heart rate, respiratory rate, oral temperature and pulse oximetry. Include scheduled time points only.


Sponsor: Insys Development Company, Inc

Table 14.3.4
Summary of Physical Exam Findings
Safety Population

| | | Standard Narcotic<br>Therapy[1] | Buprenorphine SL Spray<br>(0.5 mg TID) | Overall |
|---|---|---|---|---|
| | | N=xx | N=xx | N=xx |
| Study Visit | Exam Finding | n (%) [1] | n (%) [1] | n (%) [1] |
| Screening | n | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Normal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Abnormal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Not Done | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pre-surgery | n | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Normal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Abnormal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Not Done | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Treatment Period/ 72 h | n | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Normal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Abnormal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Not Done | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Etc. | | | | |

## Footnote:

[1] Subjects assigned Standard Narcotic Therapy were given morphine IV 4 mg TID for 24 hours, followed by Oxycodone Hydrochloride tablet, 10 mg TID for the remainder of the treatment period.

# Programmer note:

Include scheduled time points only.


Sponsor: Insys Development Company, Inc

Table 14.3.5
Summary of Oral Cavity Exam Findings
Safety Population

| | | Standard Narcotic | Buprenorphine SL Spray | Overall |
|---|---|---|---|---|
| | | Therapy[2] | (0.5 mg TID) | |
| | | N=xx [1] | N=xx [1] | N=xx [1] |
| Study Visit/ | | | | |
| Time point [1] | Exam Finding | n (%) | n (%) | n (%) |
| Screening | n | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Screening | Active Infection | | | |
| | | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Mucositis | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Cold Sores | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Decemb Has Decembed | VV (VV V0) | VV (VV VO) | VV (VV V0.) |
| | Recent Hx Dental | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Disease | | | |
| | Other | | | |
| Pre-surgery | n | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Active Infection | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Mucositis | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Cold Sores | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pre-dose | n | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Active Infection | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Mucositis | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Cold Sores | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Etc. | | | | |

#### Footnote:

# Programmer note:

Include scheduled time points only.

<sup>[1]</sup> During treatment period, oral cavity exam will be performed at 90 min, 12h, 24h, 48h, and 72h after dosing.

<sup>[2]</sup> Subjects assigned Standard Narcotic Therapy were given morphine IV 4 mg TID for 24 hours, followed by Oxycodone Hydrochloride tablet, 10 mg TID for the remainder of the treatment period.


Sponsor: Insys Development Company, Inc

Table 14.3.6
Summary of ECG Exam Findings
Safety Population

| | | Standard Narcotic | Buprenorphine SL | Overall |
|---|---|---|---|---|
| | | Therapy[2] | Spray (0.5 mg TID) | |
| | ECG Findings | N = xx | N = xx | N = xx |
| Study Visit / Time Points [1] | | | | |
| Screening | n | X.X (X.XX) | X.X (X.XX) | X.X (X.XX) |
| | Normal | X.X (X.XX) | X.X (X.XX) | X.X (X.XX) |
| | Abnormal | X.X (X.XX) | X.X (X.XX) | X.X (X.XX) |
| | Not Done | X.X (X.XX) | X.X (X.XX) | X.X (X.XX) |
| Pre-dose | n | X.X (X.XX) | X.X (X.XX) | X.X (X.XX) |
| | Normal | X.X (X.XX) | X.X (X.XX) | X.X (X.XX) |
| | Abnormal | X.X (X.XX) | X.X (X.XX) | X.X (X.XX) |
| | Not Done | X.X (X.XX) | X.X (X.XX) | X.X (X.XX) |
| Treatment Period / 90 min | n | X.X (X.XX) | X.X (X.XX) | X.X (X.XX) |
| | Normal | X.X (X.XX) | X.X (X.XX) | X.X (X.XX) |
| | Abnormal | X.X (X.XX) | X.X (X.XX) | X.X (X.XX) |
| | Not Done | X.X (X.XX) | X.X (X.XX) | X.X (X.XX) |
| Etc. | | | | |

#### Footnotes:

# Programmer note:

Include scheduled time points only.

<sup>[1]</sup> During treatment period, ECG exam will be performed at 90 min, 12h, 24h, 48h, and 72h after dosing.

<sup>[2]</sup> Subjects assigned Standard Narcotic Therapy were given morphine IV 4 mg TID for 24 hours, followed by Oxycodone Hydrochloride tablet, 10 mg TID for the remainder of the treatment period.


Table 14.3.7

Summary of ECG Results and Changes from Baseline by Study Visit

Safety Population

| HR (beats/min) (for example) | | | | | | |
|---|---|---|---|---|---|---|
| | Standard Narcotic Therapy[2] N=XX | | Buprenorphine SL Spray (0.5 mg TID) N=XX | | Overall<br>N=XX | |
| Study Visit/ Time point [1] Statistic | Actual | Change From<br>Baseline | Actual | Change From<br>Baseline | Actual | Change From<br>Baseline |
| Screening (Baseline) n Mean (S.D.) Median Range (Min, Max) | XXX<br>XX.X (XX.XX)<br>XXX<br>(XXX, XXX) | | XXX<br>XX.X (XX.XX)<br>XXX<br>(XXX, XXX) | | XXX<br>XX.X (XX.XX)<br>XXX<br>(XXX, XXX) | |
| 90 min<br>n<br>Mean (S.D.))<br>Median<br>Range (Min, Max) | XXX<br>XX.X (XX.XX)<br>XXX<br>(XXX, XXX) | XXX<br>XX.X (XX.XX)<br>XXX<br>(XXX, XXX) | XXX<br>XX.X (XX.XX)<br>XXX<br>(XXX, XXX) | XXX<br>XX.X (XX.XX)<br>XXX<br>(XXX, XXX) | XXX<br>XX.X (XX.XX)<br>XXX<br>(XXX, XXX) | XXX<br>XX.X (XX.XX)<br>XXX<br>(XXX, XXX) |
| Etc n Mean (S.D.)) Median Range (Min, Max) | XXX<br>XX.X (XX.XX)<br>XXX<br>(XXX, XXX) | XXX<br>XX.X (XX.XX)<br>XXX<br>(XXX, XXX) | XXX<br>XX.X (XX.XX)<br>XXX<br>(XXX, XXX) | XXX<br>XX.X (XX.XX)<br>XXX<br>(XXX, XXX) | XXX<br>XX.X (XX.XX)<br>XXX<br>(XXX, XXX) | XXX<br>XX.X (XX.XX)<br>XXX<br>(XXX, XXX) |
| Etc. | | | | | | |

<sup>[1]</sup> During treatment period, ECG exam will be performed at 90 min, 12h, 24h, 48h, and 72h after dosing Footnotes:

<sup>[2]</sup> Subjects assigned Standard Narcotic Therapy were given morphine IV 4 mg TID for 24 hours, followed by Oxycodone Hydrochloride tablet, 10 mg TID for the remainder of the treatment period.


Sponsor: Insys Development Company, Inc

# 14.1 FIGURE SPECIFICATIONS

Figure 14.1
Time To First Use Of Rescue Medication
Safety Population



Footnote:

If a subject does not take rescue medication for nausea but prematurely discontinues from the study, then the subject will be censored at the time of discontinuation. If a subject never takes rescue medication for nausea and completes the treatment phase of the study, then the subject will be considered censored at 7 days.

Points on graph represent censored events.


Sponsor: Insys Development Company, Inc

# **14.2 LISTING SPECIFICATIONS**

Sponsor: Insys Development Company, Inc

# Listing 16.2.1.1 Subject Enrollment and Randomization All Subjects

| ИММуууу ddMMM | yyyy ddMMMyyyy | 37 | | | | |
|---|---|---|---|---|---|---|
| | 1111 (00:11:1111 | Yes | ddMMMyyyy<br>(hh:mm) | XXXX | Buphrenorphine SL Spray (0.5 mg TID) | Yes/No |
| MMyyyy ddMMMy | уууу ddMMMуууу | No | | | | |
| MMyyyy ddmmm | уууу ddMMMуууу | Yes | ddMMMyyyy<br>(hh:mm) | XXXX | Standard<br>Narcotic<br>Therapy | Yes/No |
| | | | | Mуууу ddMMMуууу Yes ddMMMуууу | Mуууу ddMMMуууу ddMMMуууу Yes ddMMMуууу XXXX | Myyyy ddMMMyyyy ddMMMyyyy Yes ddMMMyyyy XXXX Standard (hh:mm) Narcotic |


Sponsor: Insys Development Company, Inc

## Listing 16.2.1.3 Subject Disposition All Subjects

Treatment: Buprenorphine SL Spray (0.5 mg TID)

| Site-Subject | End of Study<br>status [1] | Date of Last Study Visit (Study Day[2]) | Date of<br>Last<br>Subject<br>Contact | Primary Reason for Early Termination [3] | If AE<br>Specify AE<br># | If Protocol<br>Deviation,<br>Specify # | If Death,<br>Specify<br>Date | If Other -<br>Specify |
|---|---|---|---|---|---|---|---|---|
| XXX-XXX | XXXXXX | ddMMMyyyy<br>(xx) | ddMMMyyyy | XXXXXX | XX | XX | ddMMMyyyy | XXXXXXX |
| XXX-XXX | XXXXXX | ddMMMyyyy | ddMMMyyyy | XXXXXX | XX | XX | ddMMMyyyy | XXXXXXX |
| XXX-XXX<br>Etc. | XXXXXX | ddMMMyyyy | ddMMMyyyy | XXXXXXX | XX | XX | ddMMMyyyy | XXXXXXX |

- [1] End of study status can be: Study completer, Early termination.
- [2] Study Day = Date of Last Visit Date of First Treatment + 1.
- [3] Primary Reason for Early Termination can be: Adverse event (specify AE #), Death (specify date), Lost to follow-up, Protocol Violation (specify deviation #), Withdrawal of Consent by Subject, Subject Noncompliance, Study Enrollment Stopped, Other (Specify).


Sponsor: Insys Development Company, Inc

## Listing 16.2.2.1 Protocol Deviations Safety Population

Treatment: Buprenorphine SL Spray (0.5 mg TID)

| Site-Subject | Any | Deviation | Date of | Deviation | Deviation Description | Major Deviation? |
|---|---|---|---|---|---|---|
| | Deviation? | Number | Deviation | Category | | |
| | | | | [1] | | |
| XXX-XXX | Yes/No/NA | XX | ddMMMyyyy | XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Yes/No |
| XXX-XXX | Yes/No/NA | XX | ddMMMyyyy | XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Yes/No |
| XXX-XXX | Yes/No/NA | XX | ddMMMyyyy | XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Yes/No |
| Etc. | | XX | | | | |

<sup>[1]</sup> Deviation category can be: Informed consent procedure, inclusion/exclusion criteria, study medication, prohibited medications, study procedures, visit or assessment time window, missed visit or assessment, other.


Sponsor: Insys Development Company, Inc

# Listing 16.2.4.1 Demographics and Baseline Characteristics Safety Population

Treatment: Buprenorphine SL Spray (0.5 mg TID)

| Site-Subject | Date of Birth | Age (yrs)<br>[1] | Sex | Race [2] | Ethnicity<br>[3] | Baseline<br>PONV Score<br>[4]<br>/Category | Baseline<br>Height<br>(cm) | Baseline<br>Weight<br>(kg) | Baseline<br>BMI (kg/m2) |
|---|---|---|---|---|---|---|---|---|---|
| XXX-XXX | ddMMMyyyy | XX | M/F | XXXXX | XXXXX | X /Low Risk | XXX | XX.X | XX.X |
| XXX-XXX | ddMMMyyyy | XX | M/F | XXXXX | XXXXX | X /High<br>Risk | XXX | XX.X | XX.X |
| XXX-XXX<br>Etc. | ddMMMyyyy | XX | M/F | XXXXX | XXXXX | X | XXX | XX.X | XX.X |

- [1] Age is calculated at date of Informed Consent.
- [2] Race can be: White, Black or African American, Asian, American Indian or Alaskan Native, Native Hawaiian or Other Pacific Islander, or Other.
- [3] Ethnicity can be: Hispanic or Latino or Not Hispanic or Latino.
- [4] PONV score can be from 0 to 4, Scores of 0-2 are categorized as Low Risk, Scores of 3-4 are categorized as High Risk.


Sponsor: Insys Development Company, Inc

## Listing 16.2.4.2 Medical/Surgical History Safety Population

Treatment: Buprenorphine SL Spray (0.5 mg TID)

| Site-Subject | Any | HX Number | Diagnosis / Condition | System | Preferred | Start Date | Stop Date | Ongoing? |
|---|---|---|---|---|---|---|---|---|
| | Medical | | / Event | Organ | Term[1] | (Time) | (Time) | |
| | Hx? | | | Class[1] | | | | |
| XXX-XXX | Yes/No | XX | XXXXXXXXX | XXXXXXXXX | XXXXXXXXX | ddMMMyyyy | ddMMMyyyy | Yes/No |
| | | | | | | (hh:mm) | (hh:mm) | |
| XXX-XXX | Yes/No | XX | XXXXXXXXX | XXXXXXXXX | XXXXXXXXX | ddMMMyyyy | ddMMMyyyy | Yes/No |
| | | | | | | (hh:mm) | (hh:mm) | |
| XXX-XXX | Yes/No | XX | XXXXXXXXX | XXXXXXXXX | XXXXXXXXX | ddMMMyyyy | ddMMMyyyy | Yes/No |
| | | | | | | (hh:mm) | (hh:mm) | |
| Etc. | Yes/No | XX | XXXXXXXXX | XXXXXXXXX | XXXXXXXXX | ddMMMyyyy | ddMMMyyyy | Yes/No |
| | | | | | | (hh:mm) | (hh:mm) | |

Footnotes:

[1] System Organ Class and Preferred Term are based on the Version 19.0 of the MedDRA coding dictionary.


Sponsor: Insys Development Company, Inc

Listing 16.2.4.3
Prior and Concomitant Medications
Safety Population

Treatment: Buprenorphine SL Spray (0.5 mg TID)

| Site-<br>Subject | Any<br>med<br>s? | Med # | ATC Class /<br>Pref. Term/<br>Verbatim Term | Dose /<br>Units /<br>Frequenc<br>y /<br>Route<br>[1] | Start<br>Date<br>(Time) | Stop<br>Date<br>(Time) | On-<br>going? | Prior/<br>Con-<br>comitant[3] | Category [2]/ Indication | Was<br>treatme<br>nt<br>given<br>for AE<br>or MH? | AE<br># | мн # |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX-XXX | Yes<br>/No | XX | Antithrombotic Agent/ Acetylsalicylic acid / Aspirin | 81 mg /<br>QID / PO | ddMMMyyy<br>Y<br>(hh:mm) | ddMMMyyy<br>y<br>(hh:mm) | Yes/No | P/C | Concomitant Med / Cerebrovasc ular Accident Prophylaxis | Yes/No | XX | XX |
| XXX-XXX | Yes<br>/No | XX | XXXXXXXXX /<br>XXXXXXXXX /<br>XXXXXXXXX | XX XX /<br>XXX /<br>XXX | ddMMMyyy<br>Y<br>(hh:mm) | ddMMMyyy<br>y<br>(hh:mm) | Yes/No | | | Yes/No | XX | XX |
| XXX-XXX | Yes<br>/No | XX | XXXXXXXXX /<br>XXXXXXXXX /<br>XXXXXXXXX | XX XX /<br>XXX /<br>XXX | ddMMMyyy<br>y<br>(hh:mm) | ddMMMyyy<br>y<br>(hh:mm) | Yes/No | | | Yes/No | XX | XX |
| Etc. | Yes<br>/No | XX | | | ddMMMyyy<br>y<br>(hh:mm) | ddMMMyyy<br>Y<br>(hh:mm) | Yes/No | | | Yes/No | XX | XX |

### Footnote:

[1] Unit can be: Mg, mcg, ml, Capsule, Tablet, or Other. Route can be: Oral, Inhalation, Topical, IV, IM, Other. Frequency can be: QD, BID, TID, QID, Once, PRN, or Other.

- [2] Category can be: Prior Medication, Concomitant Medication, or Prophylaxis.
- [3] Prior medications are those that stop prior to the start of the first study drug administration. Any medication that stops at or after the start of the first study drug administration or with missing stop dates is considered a concomitant medication.


Sponsor: Insys Development Company, Inc

Listing 16.2.4.4 Non-Medication Therapy Safety Population

Treatment: Buprenorphine SL Spray (0.5 mg TID)

| Site-Subject | Any | Ther | ATC Class / | Dose / | Indicatio | Start | Stop | On- | Prior/ | Was | A | М |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Thera | apy | Pref. Term/ | Units / | n | Date | Date | going? | Concomitan | treatmen | E | H |
| | py? | Numb | Rescue | Frequenc | | (Time) | (Time) | | t[1] | t given | # | # |
| | | er | Medication | у / | | | | | | for AE | | |
| | | | Name | Route | | | | | | or MH? | | |
| XXX-XXX | Yes/N | Χ | XXXXXXXXX / | 81 mg / | XXXXXXXXX | ddMMMyyy | ddMMMyyy | Yes/No | P/C | Yes/No | Х | Χ |
| | 0 | | XXXXXXXXX / | QID / PO | | У | У | | | | X | X |
| | | | XXXXXXXXX | | | (hh:mm) | (hh:mm) | | | | | |
| XXX-XXX | Yes/N | X | XXXXXXXXX / | XX XX / | XXXXXXXX | ddMMMyyy | ddMMMyyy | Yes/No | | Yes/No | Х | X |
| | 0 | | XXXXXXXXX / | XXX / | | У | У | | | | Х | X |
| | | | XXXXXXXXX | XXX | | (hh:mm) | (hh:mm) | | | | | |
| XXX-XXX | Yes/N | X | XXXXXXXXX / | XX XX / | XXXXXXXX | ddMMMyyy | ddMMMyyy | Yes/No | | Yes/No | Х | X |
| | 0 | | XXXXXXXXX / | XXX / | | У | У | | | | Х | X |
| | | | XXXXXXXXX | XXX | | (hh:mm) | (hh:mm) | | | | | |
| Etc. | Yes/N | X | XXXXXXXXX / | XX XX / | XXXXXXXX | ddMMMyyy | ddMMMyyy | Yes/No | | Yes/No | Χ | X |
| | 0 | | XXXXXXXXX / | XXX / | | У | У | | | | Χ | X |
| | | | XXXXXXXXX | XXX | | (hh:mm) | (hh:mm) | | | | | |

Footnote:

[1] Prior therapies are those that stop prior to the start of the first study drug administration. Any therapy that stops at or after the start of the first study drug administration or with missing stop dates is considered a concomitant therapy.


Sponsor: Insys Development Company, Inc

Listing 16.2.4.5
Serology Laboratory And Pregnancy Test Results
Safety Population

Treatment: Buprenorphine SL Spray (0.5 mg TID)

| Site-Subject | Age | Sex | If Female, Is Subject<br>of Child Bearing<br>Potential? | Test Performed | Study Visit | Date (Time) | Result |
|---|---|---|---|---|---|---|---|
| XXX-XXX | XX | M/F | Yes/No | HIV Test Results | Screening | ddMMMyyyy (HH:MM) | Negative/Positive |
| XXX-XXX | XX | M/F | Yes/No | Hep B Antigen Results | Screening | ddMMMyyyy (HH:MM) | Negative/Positive |
| XXX-XXX | XX | M/F | Yes/No | Hep C Antigen Results | Screening | ddMMMyyyy (HH:MM) | Negative/Positive |
| XXX-XXX | XX | M/F | Yes/No | Serum Pregnancy | Screening | ddMMMyyyy (HH:MM) | Negative/Positive |
| XXX-XXX | XX | M/F | Yes/No | Urine Pregnancy | Pre-Surgery | ddMMMyyyy (HH:MM) | _ |
| XXX-XXX | XX | M/F | Yes/No | HIV Test Results | Screening | ddMMMyyyy (HH:MM) | |
| Etc. | | | | | | | |


Sponsor: Insys Development Company, Inc

# Listing 16.2.4.6 Alcohol Breath Test and Urine Drug Screen[1] Safety Population

Treatment: Buprenorphine SL Spray (0.5 mg TID)

| Site-Subject | Test performed? | Study Visit | Was Test | Date (Time) | Result |
|---|---|---|---|---|---|
| | | | Performed? | • | |
| XXX-XXX | Alcohol Test | Screening | Y | ddMMMyyyy (HH:MM) | Negative/Positive |
| XXX-XXX | | Day 1 | Y | ddMMMyyyy (HH:MM) | Negative/Positive |
| XXX-XXX | Urine Drug Screen | Screening | Y | ddMMMyyyy (HH:MM) | Negative/Positive |
| Etc. | | Day 1 | N | | |

### Footnote:

[1] Screened Drugs Found can be: Amphetamines, Barbiturates, Benzodiazepines, Cocaine, Marijuana, Methadone, Methamphetamines, Opiates, Oxycodone, Phencyclidine (PCP) Tricyclic antidepressant, or Methylenedioxymethamphetamine, Other.


Sponsor: Insys Development Company, Inc

Listing 16.2.4.7 Surgery Safety Population

Treatment: Buprenorphine SL Spray (0.5 mg TID)

| Site-Subject | Surgical Procedure [1] | Target foot for | Breast Implant | Date | Start Time | Stop Time |
|---|---|---|---|---|---|---|
| | | Bunionectomy | Size: Left/Right | | | |
| XXX-XXX | XXXXXXX | | ххх / ууу | ddMMMyyyy | hh:mm | hh:mm |
| XXX-XXX | XXXXXXX | Left | | ddMMMyyyy | hh:mm | hh:mm |
| XXX-XXX | XXXXXXX | | | ddMMMyyyy | hh:mm | hh:mm |
| Etc. | XXXXXXX | | | ddMMMyyyy | hh:mm | hh:mm |

### Foootnote:

[1] The surgical procedures will be bunionectomy, breast augmentation, or abdominoplasty.


Sponsor: Insys Development Company, Inc

## Listing 16.2.5.1 Study Drug Administration Safety Population

Treatment: Buprenorphine SL Spray (0.5 mg TID)

| Site-Subject | Study<br>Treatment<br>Period [1] | Study Medication<br>Dose [2] | Was Dose<br>Administered? | Date (Time) | If No, Specify? | Did the subject hold spray<br>under tongue for 30 sec<br>before swallowing?[3] |
|---|---|---|---|---|---|---|
| XXX-XXX | Inpatient | Dose 1 | Yes/No | ddMMMyyyy<br>(HH:MM) | XXXXXXXXX | Yes/No |
| XXX-XXX | Inpatient | Dose 2 | Yes/No | ddMMMyyyy<br>(HH:MM) | XXXXXXXXX | Yes/No |
| XXX-XXX | Inpatient | Etc. | Yes/No | ddMMMyyyy<br>(HH:MM) | XXXXXXXXX | Yes/No |
| XXX-XXX | Outpatient | Dose 1 | Yes/No | ddMMMyyyy<br>(HH:MM) | XXXXXXXXX | Yes/No |
| XXX-XXX | Outpatient | Etc. | Yes/No | ddMMMyyyy<br>(HH:MM) | XXXXXXXXX | Yes/No |
| XXX-XXX | Inpatient | Dose 1 | Yes/No | ddMMMyyyy<br>(HH:MM) | XXXXXXXXX | Yes/No |
| Etc. | | | | | | |

- [1] Study Treatment Period can be Inpatient (Days 1-4), or Outpatient (Days 4-7).
- [2] There are a possible 12 doses each for each Treatment Period.
- [3] For Buprenorphine SL Spray (0.5 mg TID) subjects only.


Sponsor: Insys Development Company, Inc

# Listing 16.2.5.2 Discharge to Outpatient Treatment Safety Population

Treatment: Buprenorphine SL Spray (0.5 mg TID)

| Site-Subject | Did subject<br>continue to<br>Outpatient | Did subject sign<br>the Opioid<br>Agreement? | Discharge Date<br>(Time) | Did subject receive<br>all Outpatient<br>instructions per | Did staff<br>dispense<br>outpatient | Did staff<br>dispense<br>study drug? |
|---|---|---|---|---|---|---|
| | Treatment | | | protocol? | diaries? | |
| XXX-XXX | Yes/No | Yes/No | ddMMMyyyy (HH;MM) | Yes/No | Yes/No | Yes/No |
| | Yes/No | Yes/No | ddMMMyyyy (HH;MM) | Yes/No | Yes/No | Yes/No |

Note:

Subjects assigned Standard Narcotic Therapy of care were given morphine IV 4 mg TID for 24 hours, followed by Oxycodone Hydrochloride tablet, 10 mg TID for the remainder of the treatment period. Subjects assigned to Buprenorphine SL Spray (0.5 mg TID) received Buprenorphine sublingual spray 0.5 mg TID for the entire treatment period. During the outpatient portion of the trial, subjects assigned to Standard Narcotic Therapy of care were instructed to take study medication only when they experienced pain, while subjects assigned to Buprenorphine SL Spray (0.5 mg TID) were instructed to maintain the TID dosing for the entire outpatient period.


Sponsor: Insys Development Company, Inc

Listing 16.2.5.3 Study Drug Accountability Safety Population

Treatment: Buprenorphine SL Spray (0.5 mg TID)

| Site-Subject | Dispensed<br>Date<br>(Time) [1] | Number of<br>study<br>devices or<br>pills<br>dispensed | Did subject return Outpatient Diaries? If No, specify reason | Date | Did the<br>subject<br>return<br>study<br>drug? | Date | Number of unused study devices or pills returned | Number of<br>used study<br>devices<br>returned | Did the subject return fewer than expected devices or pills? If Yes, was an IP irregularities form completed? |
|---|---|---|---|---|---|---|---|---|---|
| XXX-XXX | ddMMMyyyy<br>(HH;MM) | XX | Yes | ddMMMyyyy | Yes/No | ddMMMyyyy | XX | XX | Yes, Yes |
| XXX-XXX | ddMMMyyyy<br>(HH;MM) | XX | No,<br>XXXXXXX | | Yes/No | ddMMMyyyy | XX | XX | No |
| XXX-XXX | ddMMMyyyy<br>(HH;MM) | XX | Yes/No | ddMMMyyyy | Yes/No | ddMMMyyyy | XX | XX | Yes/No |

Footnote:

[1] Subjects were dispensed diaries and study drug for outpatient treatment period at the Site Discharge.


Sponsor: Insys Development Company, Inc

Listing 16.2.5.4
Rescue Medication Administration
Safety Population

Treatment: Buprenorphine SL Spray (0.5 mg TID)

| Was Rescue<br>Medication | Rescue<br>Medication # | ATC Class /<br>Pref. Term/ | Dose / Unit /<br>Route [1] | Date (Time) | Medication<br>Category |
|---|---|---|---|---|---|
| Administered? | | Rescue Medication | | | |
| | Name | | | | |
| Yes/No | 1 | XXXXXXXXX / | XXX / XXX/ XXXX | ddMMMyyyy (HH:MM) | Pain/Nausea |
| | | XXXXXXXXX / | | | |
| | | XXXXXXXXX | | | |
| Yes/No | 2 | XXXXXXXXX / | XXX / XXX/ XXXX | ddMMMyyyy (HH:MM) | Pain/Nausea |
| | | XXXXXXXXX / | | | |
| | | XXXXXXXXX | | | |
| XXX-XXX Yes/No | Etc. | XXXXXXXXX / | XXX / XXX/ XXXX | ddMMMyyyy (HH:MM) | Pain/Nausea |
| | | XXXXXXXXX / | | | |
| | | XXXXXXXXX | | | |
| Yes/No | XX | XXXXXXXXX / | XXX / XXX/ XXXX | ddMMMyyyy (HH:MM) | Pain/Nausea |
| | | XXXXXXXXX / | | | |
| | | XXXXXXXXX | | | |
| Yes/No | XX | XXXXXXXXX / | XXX / XXX/ XXXX | ddMMMyyyy (HH:MM) | Pain/Nausea |
| | | XXXXXXXXX / | | | |
| | | XXXXXXXXX | | | |
| Yes/No | XX | XXXXXXXXX / | XXX / XXX/ XXXX | ddMMMyyyy (HH:MM) | Pain/Nausea |
| | | XXXXXXXXX / | | | |
| | | XXXXXXXXX | | | |
| | Medication Administered? Yes/No Yes/No Yes/No Yes/No Yes/No | Medication # Medication # Yes/No 1 Yes/No 2 Yes/No Etc. Yes/No XX Yes/No XX | Medication Administered? Medication # Rescue Medication Name Yes/No 1 XXXXXXXXXX / XXXXXXXXX / XXXXXXXXXX / XXXXXX | Medication Administered? Medication # Rescue Medication Name Pref. Term/ Rescue Medication Name Route [1] Yes/No 1 XXXXXXXXXX / XXXX / XXXX / XXXX / XXXX XXXX XXXXXXXXXX / XXXX / XXXX / XXXX XXXX Yes/No 2 XXXXXXXXXX / XXXX / XXX / XXX / XXXX / XXXX XXXX XXX / XXX / XXX / XXX / XXXX XXX Yes/No XX XXXXXXXXXX / XXXX / XXX / XXX / XXX / XXXX / XXXX XXX / XXXXXX | Medication Administered? Medication Rescue Medication Name Route [1] Yes/No 1 XXXXXXXXXX / XXXX XXXX XXXX XXXX XXXX |

### Footnote:

[1] Route can be Oral or Intravenous.


Sponsor: Insys Development Company, Inc

# Listing 16.2.7.1 All Treatment Emergent Adverse Events (TEAEs) Safety Population

Treatment: Buprenorphine SL Spray (0.5 mg TID)

| Site-Subject | AE<br>Number | System Organ Class / Preferred Term[1] / Verbatim Term | Start Date (Time) / Stop Date (Time) / Duration | Ongoing? /<br>Outcome [2] | Causality[3]/ Severity[4]/ Action Taken[5] | Serious? / Specify Cause[6]/ SAE Outcome[7] |
|---|---|---|---|---|---|---|
| XXX-XXX | 1 | Injury, poisoning and procedural complications / Concussion / Concussion secondary to xxxx | 01Jan2013 (8:45) /<br>10Jan 2013 (9:00) /<br>10 days | No / Resolved | Not related<br>/Severe<br>/None | Yes /<br>Is Life<br>Threatening /<br>Drug Withdrawn |
| XXX-XXX | | | | | | |
| XXX-XXX | | | | | | |
| XXX-XXX | | | | | | |
| Etc. | | | | | | |

- [1] SOC and PT are determined by coding the verbatim term using the MedDRA Version 19.0 dictionary.
- [2] Outcome can be: Event Resolved, Resolved with sequelae, Ongoing, or Death. If SAE, outcome can be: Not Recovered/Not Resolved, Death or Other.
- [3] Causality can be: Definitely Related, Probably Related, Possibly Related, Unlikely Related, or Not Related.
- [4] Severity can be: Mild, Moderate, or Severe.
- [5] Action Taken can be: None, Study Drug Discontinued, Dose Modified, Required Concomitant Medication, Required Procedure, or Other.
- [6] Specify cause can be: Death, Life-threatening, In-patient hospitalization or prolongation of existing hospitalization, Persistent or significant disability or incapacity, Congenital anomaly or birth defect, is medically significant or requires intervention to prevent one of the outcomes listed above.
- [7] If SAE, action taken can be: None, Treatment, Unknown or Drug Withdrawn.


Sponsor: Insys Development Company, Inc

Non-Unique Tables

Listing 16.2.7.2
Treatment Related TEAEs
Safety Population

Listing 16.2.7.3 Serious TEAEs Safety Population

Listing 16.2.7.4
Deaths
Safety Population

Listing 16.2.7.5
TEAEs Leading To Premature Study Discontinuation
Safety Population


Sponsor: Insys Development Company, Inc

Listing 16.2.8.1.1 Chemistry Laboratory Results Safety Population

Treatment: Buprenorphine SL Spray (0.5 mg TID)

| Site-Subject | Study Visit | Date (Time) | Test[1,2] | Value | Units | Lower Limit | Upper Limit |
|---|---|---|---|---|---|---|---|
| | | | | | | of Normal | of Normal |
| XXX-XXX | Screening | ddMMMyyyy<br>(hh:mm) | Albumin | XX.X | XX | XX.X | XX.X |
| | | ddMMMyyyy<br>(hh:mm) | Alk Phos | XX.X | XX | XX.X | XX.X |
| | Follow-up | ddMMMyyyy<br>(hh:mm) | Albumin | XX.X | XX | XX.X | XX.X |
| | | | Alk Phos | XX.X | XX | XX.X | XX.X |
| | | | Etc. | XX.X | XX | XX.X | XX.X |
| XXX-XXX | Screening | ddMMMyyyy<br>(hh:mm) | Albumin | XX.X | XX | XX.X | XX.X |
| | | | Alk Phos | XX.X | XX | XX.X | XX.X |
| | | | Etc. | XX.X | XX | XX.X | XX.X |
| | Follow-up | ddMMMyyyy<br>(hh:mm) | Albumin | XX.X | XX | XX.X | XX.X |
| | | | Alk Phos | XX.X | XX | XX.X | XX.X |
| | | | Etc. | XX.X | XX | XX.X | XX.X |

<sup>[1]</sup> Laboratory parameters are listed alphabetically.

<sup>[2]</sup> Include the following tests for Serum Chemistry: albumin, total bilirubin, total protein, calcium, alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, blood urea nitrogen, cholesterol, glucose, sodium, potassium, chloride, bicarbonate, lactate dehydrogenase, uric acid, creatinine with calculated creatinine clearance (Cockcroft-Gault method).


Sponsor: Insys Development Company, Inc

## Listing 16.2.8.1.2 Hematology Laboratory Results Safety Population

Treatment: Buprenorphine SL Spray (0.5 mg TID)

| Site-Subject | Study Visit | Date | Test [1,2] | Value | Units | Lower Limit of Normal | Upper Limit of Normal |
|---|---|---|---|---|---|---|---|
| XXX-XXX | Screening | ddMMMyyyy | WBC Count | XX.X | XX | XX.X | XX.X |
| | | ddMMMyyyy | RBC Count | XX.X | XX | XX.X | XX.X |
| | | | Etc. | XX.X | XX | XX.X | XX.X |
| XXX-XXX Follow | Follow-up | ddMMMyyyy | WBC Count | XX.X | XX | XX.X | XX.X |
| | | | RBC Count | XX.X | XX | XX.X | XX.X |
| | | | Etc. | XX.X | XX | XX.X | XX.X |
| XXX-XXX | Screening | ddMMMyyyy | WBC Count | XX.X | XX | XX.X | XX.X |
| | | ddMMMyyyy | RBC Count | XX.X | XX | XX.X | XX.X |
| | | | Etc. | XX.X | XX | XX.X | XX.X |
| XXX-XXX | Follow-up | ddMMMyyyy | WBC Count | XX.X | XX | XX.X | XX.X |
| | | | RBC Count | XX.X | XX | XX.X | XX.X |
| | | | Etc. | XX.X | XX | XX.X | XX.X |

<sup>[1]</sup> Laboratory tests are listed alphabetically.

<sup>[2]</sup> Include the following tests for hematology values: hemoglobin, hematocrit, red blood cell count, red blood cell indices, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, platelet count (or estimate), and white blood cell count including differential.


Sponsor: Insys Development Company, Inc

# Listing 16.2.8.1.3 Urinalysis Laboratory Results Safety Population

Treatment: Buprenorphine SL Spray (0.5 mg TID)

| Site-Subject | Study Visit | Date | Test [1,2] | Value | Units | Lower Limit | Upper Limit |
|---|---|---|---|---|---|---|---|
| | | | | | | of Normal | of Normal |
| XXX-XXX | Screening | ddMMMyyyy | Specific Gravity | XX.X | XX | XX.X | XX.X |
| | | ddMMMyyyy | рН | XX.X | XX | XX.X | XX.X |
| | | | Etc. | XX.X | XX | XX.X | XX.X |
| XXX-XXX | Follow-up | ddMMMyyyy | Specific Gravity | XX.X | XX | XX.X | XX.X |
| | | | рН | XX.X | XX | XX.X | XX.X |
| | | | Etc. | XX.X | XX | XX.X | XX.X |
| XXX-XXX | Screening | ddMMMyyyy | Specific Gravity | XX.X | XX | XX.X | XX.X |
| | | ddMMMyyyy | рН | XX.X | XX | XX.X | XX.X |
| | | | Etc. | XX.X | XX | XX.X | XX.X |
| XXX-XXX | Follow-up | ddMMMyyyy | Specific Gravity | XX.X | XX | XX.X | XX.X |
| | | | рН | XX.X | XX | XX.X | XX.X |
| | | | Etc. | XX.X | XX | XX.X | XX.X |

## Footnotes:

[1]Urinalysis tests are listed alphabetically.

[2] Include the following for urinalysis: pH, specific gravity, blood, glucose, protein, and ketones.


Sponsor: Insys Development Company, Inc

Listing 16.2.8.2 Vital Signs Safety Population

Treatment: Buprenorphine SL Spray (0.5 mg TID)

| Site-Subject | Study Visit / | Date | Height | Weight | OralTemp | Systolic | Diastolic | Pulse | Respiratory | Pulse |
|---|---|---|---|---|---|---|---|---|---|---|
| | Time Point | (Time) | (cm) | (kg) | (°C) | BP | BP (mmHg) | Rate | Rate (bpm) | Oximetry |
| | | | | _ | | (mmHg) | [1] | (bpm) | [2] | (Spo2) |
| | | | | | | [1] | | [2] | | [3] |
| XXX-XXX | XXXXXXXXX /<br>XXXXXX | ddMMMyyyy<br>(HH;MM) | XXX | XXX | XX.X | XXX | XXX | XXX | XX | XXX |
| | | ddMMMyyyy<br>(HH;MM) | XXX | XXX | XX.X | XXX | XXX | XXX | XX | XXX |

### Footnotes:

During treatment period,

- [1] Blood Pressure is measured every 4 hours after first dose.
- [2] Pulse rate and respiratory rate are measured at TO, 1h and every 2 hours after first dose.
- [3] Pulse Oximetry is measured at 90 min, 12h, 24h, 48h, and 72h after first dose.


Sponsor: Insys Development Company, Inc

# Listing 16.2.8.3.1 Physical Examinations Safety Population

Treatment: Buprenorphine SL Spray (0.5 mg TID)

| Site-Subject | Study Visit | Was the Physical Examination performed? | Date (Time) | Body System [1] | Status [2] | Clinical<br>Significance<br>[3] |
|---|---|---|---|---|---|---|
| XXX-XXX | | Yes/No | ddMMMyyyy<br>(HH:MM) | Dermatologic | XXXXX | XXX |
| XXX-XXX | | Yes/No | ddMMMyyyy<br>(HH:MM) | HEENT | XXXXX | XXX |
| XXX-XXX | | Yes/No | ddMMMyyyy<br>(HH:MM) | Etc. | | XXX |
| XXX-XXX | | Yes/No | ddMMMyyyy<br>(HH:MM) | Dermatologic | XXXXX | XXX |
| XXX-XXX | | Yes/No | ddMMMyyyy<br>(HH:MM) | HEENT | XXXXX | XXX |
| XXX-XXX | | Yes/No | ddMMMyyyy<br>(HH:MM) | Etc. | | XXX |

<sup>[1]</sup> Body System can be: HEENT, Cardiovascular, Respiratory, Gastrointestinal, Neurologic, Dermatologic, Musculoskeletal, or Other (Specify).

<sup>[2]</sup> Status can be: Normal, Abnormal, or Not Done.

<sup>[3]</sup> Clinical Significance can be: CS=Clinically Significant or NCS=Not Clinically Significant.


Sponsor: Insys Development Company, Inc

# Listing 16.2.8.3.2 Oral Cavity Examinations Safety Population

Treatment: Buprenorphine SL Spray (0.5 mg TID)

| Site-Subject | Study Visit /<br>Time Point [1] | Was the Oral Cavity<br>Examination performed? | Date (Time) | Observation [2] |
|---|---|---|---|---|
| XXX-XXX | XXXXXXXXX /<br>XXXXXX | Yes/No | ddMMMyyyy (HH:MM) | Active Infection, Tongue piercing |
| XXX-XXX | XXXXXXXXX /<br>XXXXXX | Yes/No | ddMMMyyyy (HH:MM) | xxxxxxxxxxxxxx |
| XXX-XXX | XXXXXXXXX /<br>XXXXXXX | Yes/No | ddMMMyyyy (HH:MM) | xxxxxxxxxxxxxxx |

<sup>[1]</sup> During treatment period, oral cavity exam will be performed at 90 min, 12h, 24h, 48h, and 72h after dosing.

<sup>[2]</sup> Observation can be: None, Active Infection, Mucositis, Cold Sores, Viral Lesions, Local Irritation, Periodontal Disease, Current piercings of the tongue or anywhere in the oral cavity, Evidence of prior piercings of the tongue or anywhere in the oral cavity, recent history of significant dental disease. Subjects may have multiple findings at each exam.


Sponsor: Insys Development Company, Inc

## Listing 16.2.8.4 ECG Exam Assessment Safety Population

Treatment: Buprenorphine SL Spray (0.5 mg TID)

| Site-Subject | Study Visit / Time Point [1] | Was the ECG performed? | Date (Time) | Parameter | Findings [2] | If Abnormal, Please<br>Describe Findings |
|---|---|---|---|---|---|---|
| XXX-XXX | XXXXXXXXX /<br>XXXXXXX | Yes/No | ddMMMyyyy (HH:MM) | HR | XX | |
| | | | | P-R Interval | XX | |
| | | | | Interpretation | Normal | |
| XXX-XXX | XXXXXXXXX /<br>XXXXXX | Yes/No | ddMMMyyyy (HH:MM) | HR | XX | |
| | | | | P-R Interval | XX | |
| | | | | <br>Intorprotection | Abnormal CC | VVVVVVVVV |
| | | / | | Interpretation | Abnormal-CS | XXXXXXXX |
| XXX-XXX | XXXXXXXXX /<br>XXXXXX | Yes/No | ddMMMyyyy (HH:MM) | | XX | |
| XXX-XXX | XXXXXXXX /<br>XXXXXX | Yes/No | ddMMMyyyy (HH:MM) | | XX | |

- [1] During treatment period, ECG exam will be performed at 90 min, 12h, 24h, 48h, and 72h after dosing.
- [2] Findings can be: Normal, Abnormal Clinically Significant (CS) or Abnormal Not Clinically Significant (NCS).


Sponsor: Insys Development Company, Inc

Listing 16.2.8.5 Comments Safety Population

Treatment: Buprenorphine SL Spray (0.5 mg TID)

| ilcacment. Dupiene | orburne on obray (0.0 | , mg iib) | | |
|---|---|---|---|---|
| Site-Subject | Study Visit | Date | CRF Page | Comment |
| XXX-XXX | XXXXXXXX | ddMMMyyyy | XXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXX-XXX | XXXXXXX | ddMMMyyyy | XXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXX-XXX | XXXXXXX | ddMMMyyyy | XXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| Etc. | XXXXXXX | ddMMMyyyy | XXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |